Protocol Number: CAL-USA-11 Document status: Final SAP Version 1.0



#### STATISTICAL ANALYSIS PLAN

AN ADAPTIVE PHASE I/II STUDY OF THE SAFETY OF CD4+ T LYMPHOCYTES AND CD34+ HEMATOPOIETIC STEM/PROGENITOR CELLS TRANSDUCED WITH LVsh5/C46, A DUAL ANTI-HIV GENE TRANSFER CONSTRUCT, WITH AND WITHOUT CONDITIONING WITH BUSULFAN IN HIV-1 INFECTED ADULTS PREVIOUSLY EXPOSED TO **ART** 

Protocol No.: CAL-USA-11

Product Code: Cal-1

PREPARED FOR: Calimmune Australia Pty

> Ltd: Level 8, Lowy Packer Building, 405 Liverpool Street, Darlinghurst NSW 2010,

Sydney, Australia

Calimmune, Inc.

5151 E. Broadway Blvd., Suite 700,

Tucson, AZ 85711

USA

PREPARED BY:



DATE OF ISSUE: 15 December 2017

VERSION/STATUS: Draft Version 1.0 (16 June 2017)

**Draft Version 2.0 (21 July 2017)** 

Final Draft Version 1.0 (21 September 2017) Final Draft Version 2.0 (22 September 2017) Final Draft Version 3.0 (26 September 2017) Final Draft Version 4.0 (25 October 2017) Final Draft Version 5.0 (07 December 2017)

Final Version 1.0 (15 December 2017)

15 December 2017 **VERSION DATE:** 

**AUTHOR:** PPD

Document status: Final SAP Version 1.0

# SAPAPPROVAL

By my signature, I confirm that this statistical analysis plan (SAP) has been approved for use on the CAL-USA-11 study:

| Name | Title / Company | Signature | Date |
|-------------|--------------------|-----------|-----------|
| PPD | | | |
| *E-mail and | proval sent by PPD | -44 | 17:46 PST |


# Table of contents

| List of Abbreviations | 5 |
|-------------------------------------------------------------------|----|
| 1. Introduction | 7 |
| 2. Project Overview | 8 |
| 2.1. Description of Overall Study Design and Plan | 8 |
| 2.2. Objectives | 8 |
| 2.3. Sample Size | 9 |
| 2.4. Randomization and Assignment of Subjects to Treatment Groups | 10 |
| 3. Statistical Considerations | 11 |
| 4. Analysis Populations | 13 |
| 4.1. Population Descriptions | 13 |
| 5. Subject Disposition | 14 |
| 5.1. Subject disposition | 14 |
| 6. Protocol Deviations | 15 |
| 7. Demographic and Baseline Information | 16 |
| 7.1. Demographics | 16 |
| 7.2. HIV-1 history | 16 |
| 7.3. Medical history | 16 |
| 7.4. Eligibility | 16 |
| 7.5. Chest X-Ray | 16 |
| 7.6. ART Therapy History | 16 |
| 8. Study Drug Administration | 17 |
| 8.1. Transduced CD4+ and CD34+ Cell Product Dose | 17 |
| 8.2. CD4+ and CD34+ Apheresis | 17 |
| 8.3. CD4+ and CD34+ Manufacturing | 17 |
| 8.4. Mobilization Therapy | 17 |
| 8.5. Busulfan Administration and PK Data | 17 |
| 9. Pharmacokinetics | 18 |
| 10. Pharmacodynamics (PD) | 19 |
| 11. Efficacy | 20 |
| 11.1. Cell Dose vs. Marking/Expression | 20 |


| 11.2. Busulfan AUC (Cohorts 2 and 3) vs. Marking/Expression | 21 |
|---|---|
| 11.3. CD4+ and HIV-1RNA vs. Marking/Expression | 21 |
| 11.4. Absolute Neutrophil Counts (ANC) and Platelets vs. Marking/Expression | 21 |
| 11.5. Lymphocyte Development and Chronic Inflammation vs. Marking/Expression | 22 |
| 12. Safety | 23 |
| 12.1. Adverse Events | 23 |
| 12.2. Concomitant medication | 23 |
| 12.3. Laboratory | 23 |
| 12.4. Vital Signs | 24 |
| 12.5. Physical Examination | 24 |
| 12.6. Pregnancy Test | 24 |
| 12.7. Other Safety | 24 |
| 13. Immunogenicity Endpoints | 25 |
| 14. Handling of Missing Data | 26 |
| 15. Changes to the Planned Analysis | 27 |
| 16. Interim and Final Analysis | 28 |
| 16.1. Medical Review Committee (MRC) | 28 |
| 16.2. Data Safety Monitoring Board (DSMB) Analyses | 28 |
| 16.3. Interim Analyses | 29 |
| 16.4. Final Analysis (End of Study) | 29 |
| 17. Software | 30 |
| 18. Tables | 31 |
| 19. Listings | 32 |
| 20. Figures | 34 |
| 21. References | 36 |
| 22. Appendix I: Summary of Protocol Changes | 37 |

Protocol Number: CAL-USA-11 Document status: Final SAP Version 1.0

# **List of Abbreviations**

| Term | Abbreviation |
|---|---|
| AE | Adverse Event |
| ANC | Absolute Neutrophil Count |
| ART | Antiretroviral Therapy |
| AUC | Area Under the Curve |
| Cal-1 | LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct |
| CI | Confidence Interval |
| CSR | Clinical Study Report |
| DBP | Diastolic Blood Pressure |
| DSMB | Data Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| GALT | Gut-associated Lymphoid Tissue |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte Colony-stimulating Factor |
| Н | High |
| HIV-1 | Human Immunodeficiency Virus Type 1 |
| HSPC | CD34+ Hematopoietic stem/progenitor cells |
| HSPC <sup>tn</sup> | Cal-1 transduced CD34+ Hematopoietic stem/progenitor cells |
| IP | Investigational Product |
| L | Low |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRC | Medical Review Committee |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| RCL | Replication Competent Lentivirus |
| RNA | Ribonucleic Acid |
| SAP | Statistical Analysis Plan |


| Term | Abbreviation |
|-----------------|---------------------------------------------------|
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis System |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| SUSAR | Serious and Unexpected Suspected Adverse Reaction |
| T <sup>tn</sup> | Cal-1 transduced CD4+ T lymphocytes |
| WBC | White Blood Cell |


### 1.Introduction

The following SAP provides the outline for the statistical analysis of the data from the CAL-USA-11 study (protocol version 8 dated 08 July 2015).

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post hoc analyses not necessarily identified in this SAP may be performed to further examine study data. Any post hoc, or unplanned, exploratory analyses performed will be clearly identified as such in the final CSR.


# 2. Project Overview

# 2.1.Description of Overall Study Design and Plan

# Study Design Overview:

This is an adaptive design study to evaluate the safety and feasibility of LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct (Cal-1) transduced CD34+ Hematopoietic stem/progenitor cells (HSPC) and CD4+ T lymphocytes in Human Immunodeficiency Virus Type 1 (HIV-1) infected subjects who have previously been exposed to Antiretroviral Therapy (ART) but are not currently taking any antiretroviral agent. Three cohorts of at least 3 subjects each will be enrolled:

- Cohort 1: No busulfan conditioning
- Cohort 2: Conditioning with a single dose of 4mg/kg busulfan.
- Cohort 3: Conditioning with two doses of busulfan, with first dose of 4, 3 or 2 mg/kg and second dose based on real-time pharmacokinetic-guided dosing to reach targeted drug exposure area under the curve (AUC).

Progressive enrollment of Cohort 1, then Cohort 2 and then Cohort 3 is dependent on the recommendation of an independent Data Safety Monitoring Board (DSMB).

Subjects will have cell collection procedures (aphereses) performed; first to collect unstimulated CD4+ T lymphocytes, followed by CD34+ HSPC after mobilization. The mononuclear cell populations obtained from each of these collection procedures will be separated into purified CD4+ T lymphocytes and CD34+ HSPC, respectively and processed (transduced, cultured and cryopreserved) separately.

The primary endpoint for all subjects will be at 48 weeks' post-infusion, after which they may continue follow-up for up to one additional year in the Follow-up Extension phase. All subjects will transfer to a separate long-term follow-up protocol that will monitor each subject for potential long term adverse effects of Cal-1. Secondary data points are collected up to study completion or until early withdrawal or secondary analysis endpoint criteria is met (discontinuation), whichever occurs first. Subjects should commence ART at any time during the study if CD4+ T lymphocyte counts are confirmed to decline < 350 cells/µl (mm3) and/or to less than 1/3 of the CD4+ T cell % at the defined assessment in section 3, if plasma HIV-1 RNA exceeds 250,000 copies/µl or > 20-fold increase from the defined assessment, or in event of pregnancy.

#### 2.2.Objectives

# 2.2.1.Primary objective

The primary objectives are to evaluate in HIV-1 infected adults who have previously been on ART:

- The safety and feasibility of the introduction of Cal-1, gene-transduced, hematopoietic cell populations.
- The safety of intravenous busulfan to improve HSPC<sup>tn</sup> engraftment

Safety outcomes up to study completion will be measured per the safety evaluations. Feasibility measures will include the analysis of the Cal-1 transduced CD4+ T lymphocytes (Ttn) and Cal-1 transduced CD34+ Hematopoietic stem/progenitor cells (HSPCtn) cells release criteria and characterization. Feasibility measures will include the number of T<sup>tn</sup>


and HSPC<sup>tn</sup> manufacturing procedures successfully completed (i.e. complying with all release criteria), CD4+ and CD34+ purity, expression of various surface markers, and the number of target cells harvested.

# 2.2.2.Secondary objective(s)

The secondary objectives of the study are to assess the difference between the 3 treatment cohorts in:

- The extent of HSPC<sup>tn</sup> contribution to hematopoiesis and T<sup>tn</sup> survival by evaluation of Cal-1 marking and expression in peripheral blood at time points up to study completion or discontinuation.
- The extent of HSPC<sup>tn</sup> contribution to hematopoiesis and T<sup>tn</sup> survival by evaluation of Cal-1 marking and expression in gut-associated lymphoid tissue (GALT).
- The potential benefit of busulfan conditioning as determined by;
  - o The extent of engraftment and differentiation of HSPCtn over time by evaluation of Cal-1 marking and expression in peripheral blood subpopulations (monocytes, granulocytes, CD4+ and CD8+ lymphocytes)
  - o The extent of HSPCtn engraftment by evaluation of Cal-1 marking and expression in bone marrow at Week 12, 24, 48 and early discontinuation.
- The potential efficacy of Cal-1 in controlling HIV-1 infection for each subject, as measured by;
  - o Plasma HIV-1 RNA relative to the Assessment for Comparison (as defined in section 3).
  - Plasma HIV-1 RNA over time
  - o CD4+ T lymphocyte count, percentage and CD4+/CD8+ T lymphocyte ratio relative to the Assessment for Comparison (as defined in section 3).
  - o CD4+ T lymphocyte count, percentage and CD4+/CD8+ T lymphocyte ratio over time
  - Time to commencement of ART

The endpoint for these secondary analyses is study completion, withdrawal, or until discontinuation due to secondary analysis endpoint criteria.

- Impact on lymphocyte development for each subject, as measured by changes in thymopoiesis and maturation markers (Absolute and % Total Recent Thymic Emigrant) in peripheral blood relative to the Assessment for Comparison (as defined in section 3). and impact on chronic inflammation for each subject as measured by changes in inflammation markers (%CD4+ HLA-DR+ and Total CD4+ HLA-DR+2) in peripheral blood relative to the Assessment for Comparison (as defined in section 3) over time.
- A tropism shift from R5 to dual/mixed or X4 at any time point post-infusion.

#### 2.3. Sample Size

This is a phase I/II study, and the sample size has not been based on formal power considerations. No recruitment limit is set for any of the participating sites, with the only restriction being consecutive enrollment that does not exceed 4 subjects per cohort.


Subjects in Cohorts 2 and 3 will not receive busulfan or be infused until the DSMB recommendations are received.

In terms of safety data, pooling all subjects across the three arms, the study will have at least an 80% probability of observing one or more serious adverse events if the true rate of these events in a subject is 12.6% or higher for 12 subjects, or ≥ 16.4% if 9 or more subjects. Pooling the busulfan subjects will give at least an 80% probability of observing one or more serious adverse events that occur with a true rate of 18.2% per subject for n=8, and 23.5% for n=6. Within any arm of four subjects, the study will have 80% probability of detecting events with a true rate of 33.1% per subject.

Hence the study will be well powered to detect only serious adverse events that occur with a reasonably high probability. The study will not be well powered to detect events that are rarer than about 10-20% per subject.

### 2.4.Randomization and Assignment of Subjects to Treatment Groups

This trial will not be randomized. Subjects will be consecutively enrolled into cohorts and each cohort will not exceed 4 subjects.


### 3. Statistical Considerations

Data will be handled and processed per the sponsor's representative (CCI ) Standard Operating Procedures (SOPs), which are written based on the principles of good clinical practice (GCP).

All data collected on the electronic case report forms (eCRFs) will be presented in the data sorted by cohort, subject number and visit, where applicable. All summaries will present the data by cohort, and overall (total subjects), as applicable.

Unless otherwise stated, the following statistical approaches will be taken:

- <u>Continuous variables</u>: Descriptive statistics will include the number of non-missing values (N), mean, standard deviation (SD), median, minimum, maximum.
- <u>Categorical variables</u>: Descriptive statistics will include frequency counts and percentages per category. Percentages will be rounded to one decimal place, with the denominator being the number of subjects in the relevant population with non-missing data, unless otherwise specified.
- Imputation: No missing data will be imputed.
- <u>Confidence intervals (CIs)</u>: CIs will be two-sided and will use 95% confidence levels, unless otherwise specified.
- Repeat assessments (Safety): On occasion, when the initial assessment does not yield
  a valid value), repeat assessments may be included in summary presentations (Tables,
  Figures). Original values will be used in summary presentations, unless otherwise
  noted. All assessments captured in the Electronic Data Capture (EDC) system will be
  presented in the data listings.
- <u>Correlation coefficients:</u> Pearson's product-moment correlation and Spearman's correlation coefficient will both be produced for all correlation analyses.
- One Sample t-tests: Student t-test and the signed rank test (non-parametric) will be used to calculate whether the change from assessment for comparison (as defined in section 3) in log<sub>10</sub> plasma HIV-1 RNA and CD4 count is 0 at peak CD4/HIV-RNA and Week 48. P-values and 95% CIs for the mean and median change will be presented.
- Assessments for Comparison:
  - Cal1-Marking/Expression: All data will be compared to the pre-infusion value for Cohort 1 or the pre-busulfan value for Cohorts 2 & 3.
  - CD4+ Count and HIV-1-RNA will be compared with Screening (average of Screening 1 and Screening 2 values), the final pre-Apheresis visit, and preinfusion (Cohort 1) / pre-busulfan (Cohorts 2 and 3).
  - ANC and Platelets will be compared with Screening (average of Screening 1 and Screening 2 values), the final pre-Apheresis visit, and the pre-infusion (Cohort 1) / pre-busulfan (Cohorts 2 and 3) visit.
  - CD3/CD4, CD3/CD8. CD4:CD8 ratio will be compared with Screening (average of Screening 1 and Screening 2 values), the final pre-Apheresis visit, and the pre-infusion (Cohort 1) / pre-busulfan (Cohorts 2 & 3) visit.
  - log<sub>10</sub>HIV-1 Ribonucleic acid (RNA) (Abbott and Roche assays) will be compared with Screening (average of Screening 1 and Screening 2 values), the final pre-Apheresis visit, and the pre-infusion (Cohort 1) / pre-busulfan (Cohorts 2 & 3) visit.


Peak marking/expression data: Peak marking/expression data is the maximum data value post the start of the transduced cell infusion.

- Week 48 Assessment data: The week 48 assessment data will be the data collected at the Week 48 visit, or the last visit with recorded data prior to the Week 48 visit if no data is available at the Week 48 visit.
- Cell dose will be defined as follows:
  - o CD4+: Total Number of CD4+ Cells (unit is x108) divided by weight, then converted to x10<sup>6</sup>, and finally rounded to two decimal places.
  - o CD34+: Total Number of CD34+ Cells (unit is x108) divided by weight, then converted to x10<sup>6</sup>, and finally rounded to two decimal places.

For all marking/expression data, if a "Not Detectable Value" is recorded, the value will be set to 0 for analysis purposes.

In the summary tables and figures, treatment groups will be summarized separately for each dose cohort and overall (all subjects).


# 4. Analysis Populations

Two analysis populations are defined for this study, the Enrolled and the Safety populations. Data for Screen Failures will not be included in any summary tables, figures, or data listings.

Furthermore, any additional analysis populations not identified in the SAP will be identified in the final CSR as post hoc analyses. This may include the addition of additional study populations or subgroups of interest.

The analysis population each subject is included in will be listed.

### 4.1.Population Descriptions

### 4.1.1. Enrolled Population

All Subjects enrolled who have signed informed consent will be included in the enrolled population. Screening failures will not form part of this population. Subjects who are eligible but discontinue the trial before starting the intervention phase will only form part of the enrolled population.

# 4.1.2. Safety Population

The safety population will include all enrolled subjects have signed informed consent who started the interventional phase of the trial (i.e. CD4+ Apheresis).


# **5.Subject Disposition**

# 5.1. Subject disposition

All subjects who provide informed consent (signed) and enrolled will be accounted for in this study. Subject disposition will be listed.

By-subject data listings for subject disposition will be generated, including informed consent date, study status (Ongoing, Discontinuation, Withdrawal or Completion), date of discontinuation, withdrawal or completion, reason for discontinuation or withdrawal, last schedule visit attended and inclusion into the enrolled and safety populations.

The time to starting ART from CD4+ Apheresis start will be summarized using Kaplan-Meier plots. If no antiretroviral treatment is commenced, the time period will be censored on the date of study completion/discontinuation.

The calculation will be done as follows: Date Antiretroviral Therapy Commenced / Date of Discontinuation, Withdrawal or Completion - CD4+ Apheresis Date + 1.


### **6.Protocol Deviations**

Unless there is a safety concern, there should be no deviations or violations of the study protocol.

Overall protocol deviations (major and minor deviations combined) will be summarized by study visit by frequency counts and % of the total number of subjects per cohort.

In addition, major/minor protocol deviations reported, dependent on the number of events, will be summarized by cohort and overall by frequency counts and the % of the total deviations and/or listed for each subject in the by-subject data listings. The total number of events related to the protocol and GCP will also be represented.

Prior to database lock, all protocol deviations will be reviewed and assigned a status of Minor or Major.

Major/minor protocol deviations may include the following, depending on the timing and nature of the deviation:

- Non-compliance to study medication (i.e. subjects did not receive Investigational Product (IP) as per Clinical Study Protocol)
- Lost to follow-up (i.e. not all safety, pharmacokinetic (PK) data, efficacy data points recorded as per Clinical Study Protocol)
- Use of prohibited concomitant medication
- Violation of inclusion/exclusion criteria
- Deviation from study specific instructions
- If, for any reason, the cell infusions cannot proceed as planned, busulfan conditioning should be postponed and rescheduled for as soon as possible. A delay of up to 2 weeks will not be considered a protocol deviation


# 7. Demographic and Baseline Information

Demographic will be summarized using the Enrolled Population.

# 7.1.Demographics

Demographic data, including age, gender, race, ethnicity will be summarized by cohort and overall.

A by-subject data listing for demographic characteristics will be generated.

# 7.2.HIV-1 history

HIV-1 History (including lowest CD4+ T lymphocyte count (cells/µl) and highest plasma HIV-1 viral load (copies/mL) will be summarized by cohort and overall.

The date of HIV-1 diagnosis, lowest CD4+ T Lymphocyte count (cells/µl), the date of the, lowest CD4+ T lymphocyte count (cells/µl), highest plasma HIV-1 viral load (copies/mL) and the date of the highest plasma HIV-1 viral load (copies/mL) will be listed.

# 7.3.Medical history

Medical history will be presented in the by-subject data listings. Condition, affected body system, onset date, resolution date (ongoing) and planned treatment for the condition will be recorded.

### 7.4. Eligibility

Inclusion/exclusion eligibility criteria information, including evaluation date, criteria not met, will be listed for each subject. Eligibility will be listed for all screened subjects.

### 7.5.Chest X-Ray

Chest x-ray results will be listed by visit and cohort by subject. Abnormal chest x-ray results will be flagged.

### 7.6.ART Therapy History

History of ART therapy will be listed by subject and cohort. All drugs and associated doses will be listed per regimen. For each ART, details of each regimen (drug, start date, ongoing yes/no, stop date, reason for treatment discontinuation and lowest plasma HIV-1 viral load achieved during the regimen) will be listed.


# 8.Study Drug Administration

Study cellular product administration results will be presented using the Safety Population.

### 8.1. Transduced CD4+ and CD34+ Cell Product Dose

Transduced CD4+ and CD34+ Cell Product Dose (Transduction efficiency, viability and cell numbers for T<sup>tn</sup> and HSPC<sup>tn</sup>) data will be included in the by-subject data listings.

### 8.2.CD4+ and CD34+ Apheresis

CD4+ and CD34+ (including Granulocyte Colony-stimulating Factor (G-CSF) Day 4 & plerixafor and G-CSF Day 5) apheresis data (successful completion, filtration volume (L), number of CD4+ Lymphocytes Collected (x108 cells) and number of CD34+ Lymphocytes Collected (x10<sup>8</sup> cells) will be included in the by-subject data listings.

# 8.3.CD4+ and CD34+ Manufacturing

Feasibility measures such as the number of T<sup>tn</sup> and HSPC<sup>tn</sup> manufacturing procedures successfully completed (i.e. complying with all release criteria); number of gene modified cells, as affected by CD4+ and CD34+ purity, transduction efficiency, and viability; and the number of target cells harvested will be summarized overall.

Several associations between feasibility and safety measures and efficacy endpoints will be investigated, including:

- Associations between the number of gene-modified cells infused, peripheral blood marking and expression, plasma HIV-1 RNA, CD4+ T cell counts
- Integration profile of the T<sup>tn</sup> and HSPC<sup>tn</sup> products and observations in integration analysis of peripheral blood post infusion
- HSPC<sup>tn</sup> methylcellulose colony forming units and peripheral blood subpopulation marking

The CD4+ T Lymphocyte manufacturing and the CD34+ HSPC manufacturing process along with any deviation from the manufacturing process will be documented for each subject.

### 8.4. Mobilization Therapy

The administration of G-CSF with and without plerixafor therapy (administered yes/no, dose administered (µg/kg), total daily dose (µg), full dose administered (yes/no), date of administration will be included in the by-subject data listings.

### 8.5. Busulfan Administration and PK Data

For Cohorts 2 and 3, busulfan administration data will be listed. The listing will also be inclusive of busulfan AUC (µMol/min), concentration at steady state (ng/mL) and clearance (mL/min/Kg).

In addition, busulfan AUC and clearance data will be represented graphically. Busulfan concentrations will be plotted over time (hours post dose 1 & 2) and histograms will be created for the AUC and clearance by subject by visit.


# 9.Pharmacokinetics

Included as part of busulfan administration.


# 10.Pharmacodynamics (PD)

Not applicable to this study.


# 11.Efficacy

All efficacy summary analyses will be based on the safety population. Descriptive summaries will be presented with parameters to be correlated listed by subject by cohort by visit and overall adjacent to one another.

In addition to the descriptive statistics, Pearson's product-moment correlation and Spearman's correlation coefficient will both be produced for all correlation analyses and will be presented by cohort and overall.

Scatterplots of all correlated parameters by visit by cohort (different color markings will be used for each cohort) will also be presented on a subject level.

# 11.1.Cell Dose vs. Marking/Expression

The total number of infused CD4+ Ttn and CD34+ HSPCtn (Cell Dose) cells on Day 0 will be compared to the peak marking/expression data post transduced cell infusion and to the marking/expression at Week 48.

The marking/expression data that will be included are:

- Peripheral Blood:
  - Cal-1 Marking (WPRE gPCR) (%)
  - Cal-1 Marking (WPRE qPCR) (copies/cell)
  - Cal-1 C46 Expression (C46 RTqPCR) (relative expression)
  - Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)
- Peripheral Blood Subsets: monocytes, granulocytes, CD8+ lymphocytes, CD4+ lymphocytes):
  - Cal-1 Marking (WPRE qPCR) (copies/cell)
  - Cal-1 C46 Expression (C46 RTqPCR) (relative expression)
  - Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)
- Bone Marrow:
  - Cal-1 Marking (WPRE qPCR) (copies/cell)
  - o Cal-1 C46 Expression (C46 RTgPCR) (relative expression)
  - Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)
- GALT (Location 1 & Location 2):
  - Cal-1 Marking (WPRE qPCR) (copies/cell)
  - Cal-1 C46 Expression (C46 RTqPCR) (relative expression)
  - Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)

Cal1-Marking/Expression will be listed by cohort by visit for each subject. This will include peripheral blood, bone marrow and GALT (both locations). The Cal-1 marking/Cal-1 C46 expression/Cal-1 sh5 expression will be presented by result, quantification, quantification relative expression and quantification % (peripheral blood and subsets (including population purity %)) only.


In addition to the figures (correlations) discussed above the following figures will also be produced:

Line plot of Peripheral Blood Marking by week relative to the pre-infusion (Cohort 1) or pre-busulfan (Cohorts 2 & 3) value.

- Line plot of CD4 Marking by week relative to the pre-infusion (Cohort 1) or prebusulfan (Cohorts 2 & 3) value.
- Line plot of CD8 Marking by week relative to the pre-infusion (Cohort 1) or prebusulfan (Cohorts 2 & 3) value.

# 11.2.Busulfan AUC (Cohorts 2 and 3) vs. Marking/Expression

Busulfan AUCs on Day -2 (Cohort 2) and Days -4 and -2 (Cohort 3) will be compared to the peak marking/expression data and to the marking/expression data at Week 48.

The marking/expression data is as noted for section 11.1 above (Cell dose vs. Marking/Expression).

# 11.3.CD4+ and HIV-1RNA vs. Marking/Expression

CD4+ count and HIV-1RNA (Roche and Abbott assays) assessments to be compared as referenced in section 3 will be evaluated against the peak marking/expression data and to the marking/expression data at Week 48.

HIV-1 RNA nadir values (minimum Log10 HIV-1-RNA Roche and Abbott Assays value post the start of the transduced cell infusion) will be compared to the peak marking/expression data and to the marking/expression data at Week 48.

Further assessment of changes in CD4+ count and HIV-1 RNA (Roche and Abbott) over tine in comparison to marking/expression data, including sub-population may be performed post hoc of the final analysis.

The marking/expression data is as noted for section 11.1 above (Cell dose vs. Marking/Expression).

Changes in log<sub>10</sub> plasma HIV-1 RNA and CD4+ count will be formally compared in all subjects using one-sample t-tests at the peak value and Week 48 (Student's t-test and the Signed rank test).

Exploratory analyses of log<sub>10</sub> plasma HIV-1 RNA, lymphocytes (CD4+ T lymphocyte count, CD4+ %, CD4:CD8 ratio), measures of Cal-1 marking/expression and lymphocyte development (thymopoiesis, maturation and inflammation) may use repeated measures ANOVA techniques to explore changes in these endpoints over time, and any differences between treatment groups. These analyses are not well powered, and it is accepted they will be exploratory in nature and interpreted cautiously. This exploratory analysis will not be performed as part of this SAP.

### 11.4.Absolute Neutrophil Counts (ANC) and Platelets vs. Marking/Expression

ANC and Platelet nadir values (minimum ANC and Platelet values post the start of the transduced cell infusion) will be compared to the peak marking/expression data and to the marking/expression data at Week 48.


The marking/expression data is as noted for section 11.1 above (Cell dose vs. Marking/Expression).

For ANC and Platelets values, actual values and actual changes from the timepoints in section 3 will be presented at the timepoints noted above.

# 11.5.Lymphocyte Development and Chronic Inflammation vs. Marking/Expression

Lymphocyte development (thymopoiesis and maturation markers - Absolute and % Total Recent Thymic Emigrant in peripheral blood) and impact of chronic inflammation as measured by changes in inflammation markers in peripheral blood will be compared to the peak marking/expression data and to the marking/expression data at Week 48.

For inflammation markers, the average marker values of all timepoints (post the start of the transduced cell infusion) will be compared to the peak marking/expression data and to the marking/expression data at Week 48.

The marking/expression data is as noted for section 11.1 above (Cell dose vs. Marking/Expression).


# 12.Safety

Statistical methods for the safety analyses will be primarily descriptive in nature. Each cohort will be summarized separately and combined overall. No formal statistical comparisons will be made.

Safety endpoints include Adverse Events (AEs), clinical laboratory assessments (hematology, chemistry, lymphocyte phenotype, HIV-1 RNA), abnormal vital signs (pulse rate, systolic and diastolic blood pressure, temperature and oxygen saturation), abnormal physical examination, Cal-1 marking/expression data, (peripheral blood, bone marrow and GALT) and integration analysis (including re-test), replication competent lentivirus (RCL), HIV-1 Tropism, the use of concomitant medications and C46 Immunogenicity (Humoral and Cellular Response).

Safety endpoints will be analyzed using the safety population and will be based on actual treatment received.

#### 12.1.Adverse Events

Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®, Current), and data will be summarized by System Organ Class (SOC) and Preferred Term (PT). The number and percent of subjects reporting each AE will be summarized for each cohort and overall. A subject with two or more AEs within the same level of summarization (i.e., SOC or PT) will be counted only once in that level. Subjects will also be summarized by event severity and relationship to Cal-1 and study procedures (G-CSF, plerixafor or busulfan). Percentages will be based on the number of subjects in the safety population within each cohort and overall. The number of AEs reported will also be presented.

A by-subject AE data listing including verbatim term, MedDRA SOC and PT, severity, outcome, relationship to Cal-1, relationship to study procedures (e.g. G-CSF, plerixafor, busulfan, etc.), action taken and outcome will be provided. Separate listings will be generated for serious adverse events (SAEs), grade 3/4 events and grade 3/4 Cal-1 related and study procedures (G-CSF, plerixafor or busulfan) related events.

In addition, a listing of deaths will also be created. Date of death and autopsy findings will be included.

#### 12.2.Concomitant medication

Concomitant medications are medications taken at least once after the start of CD4+ Apheresis. Medication name, dose, unit, frequency, route, start date, stop date, indication and status (continuing) will be listed.

Medications stopped prior to Apheresis will not be considered concomitant medication but will be listed as well.

#### 12.3.Laboratory

All hematology, biochemistry, lymphocyte phenotype and HIV-1 RNA parameters will be listed by cohort for each subject.

Laboratory values will be compared to normal range of the single local laboratory and values that fall outside of the normal ranges will be flagged as: H (High) and L (Low) in the data listings and the clinical significance of the abnormal results noted.


In addition, separate listings will be created for all out of range hematology and biochemistry values.

Figures of the following will also be created:

- Line plot of post busulfan white blood cell (WBC) counts by cohort by subject over time (visit);
- Line plot of post busulfan ANC by cohort by subject over time (visit);
- Line plot of post busulfan Platelets by subject over time (visit);
- Line plot of %CD3/CD4 by cohort by subject over time (visit);
- Line plot of absolute CD3/CD4 by cohort by subject over time (visit):
- Line plot of absolute CD3/CD8 by cohort by subject over time (visit);
- Line plot of CD4:CD8 ratio by cohort by subject over time (visit);
- Line plot of HIV-1 Ribonucleic (RNA) (Abbott and Roche assays) by cohort by subject over time (visit);
- Line plot of log<sub>10</sub>HIV-1-RNA (Abbott and Roche assays) by cohort by subject over time (visit). In addition, all subjects will be presented on a single page for all cohorts to further assess the time to viral load suppression of Cal-1. Time of peripheral blood gene marking and ART recommencement will be added to the figure for each subject.

# 12.4. Vital Signs

Actual values for vital signs (Systolic Blood Pressure (SBP) (mmHg), Diastolic Blood Pressure (DBP) (mmHg), Pulse Rate (beats/min), Temperature (°C) and Oxygen Saturation (%)) will be listed by cohort by visit/timepoint for each subject.

In addition, abnormal vital sign values for all parameters will be listed by cohort by visit/timepoint for each subject. Vital sign values will be compared to normal range and values that fall outside of the normal ranges will be presented.

### 12.5.Physical Examination

Physical examination values will be listed by cohort by visit/timepoint for each subject.

Additionally, abnormal physical examination values and clinical significance associated with the abnormal values will also be presented by cohort by visit/timepoint for each subject.

# 12.6.Pregnancy Test

Pregnancy results will be listed by visit and cohort by subject. For positive pregnancy tests, further laboratory results and co-infection values will be presented.

### 12.7. Other Safety

RCL (including re-test) and HIV-1 Tropism Assay will be listed by cohort by visit for each subject. Integration analysis (including re-test values), will be listed by cohort by visit/timepoint for each subject.


# 13.Immunogenicity Endpoints

Immunogenicity endpoints will be analyzed using the safety population and will be based on actual treatment received.

C46 Immunogenicity (Humoral Response and Cellular Response) will be listed by cohort by visit for each subject.


# 14. Handling of Missing Data

Missing values will generally not be imputed for all data included in the analyses.


# 15. Changes to the Planned Analysis

Changes to the study design that occurred during the life cycle of the trial will be further described in an Appendix (Appendix 1) of the SAP detailing all protocol and design changes

15 December 2017

Protocol Number: CAL-USA-11


# 16.Interim and Final Analysis

# 16.1.Medical Review Committee (MRC)

A medical review committee will be established to ensure that the safety of subjects participating in the study is not compromised. The MRC will include, but will not be limited to, at least two expert physicians in the area of HIV medicine and/or hematology. The MRC will include members from the Sponsor and external consultants. The MRC will monitor the safety of the study by reviewing AE/SAE, clinical, and laboratory data in a regular and timely manner. Any grade three or four toxicities will be comprehensively reviewed and the MRC will be required to make formal recommendations. Specific recommendations concerning the dose of busulfan will be made by the MRC following assessment of postconditioning hematopoietic recovery. Delayed hematopoietic recovery is defined as an ANC <  $0.5 \times 10^3 / \mu L$  (mm<sup>3</sup>) and/or platelet count of <  $25 \times 10^3 / \mu L$  (mm<sup>3</sup>) after 42 days' postinfusion, and observation of this adverse event in any subject will prompt a reduction in the busulfan dose. The MRC will communicate any occurrence of delayed hematopoietic recovery to the DSMB in real-time.

The MRC will assess the hematopoietic recovery of every subject, and following completion of week 12 make formal recommendation if the back-up apheresis product is no longer required. With the agreement of the Principal Investigator, these samples may then be destroyed, or donated to research, in accordance with the subject's wishes at time of study consent.

The MRC will also be responsible for the review and/or input into the case narratives for Serious and Unexpected Suspected Adverse Reactions (SUSARs), including adjudication of possible causality to Cal-1 or study procedures.

Details of the composition, roles, responsibilities, and relationship with the DSMB are documented in the MRC charter.

### 16.2.Data Safety Monitoring Board (DSMB) Analyses

An independent DSMB will be commissioned for this study to evaluate the risk/benefit of busulfan and to review all safety and selected efficacy (such as the degree of Cal-1 marking in peripheral blood, GALT and bone marrow) data from cohorts 1 and 2 prior to proceeding with the next planned cohort. Progression to each cohort is dependent on the positive recommendation of the DSMB. Details of the composition, roles, responsibilities and timelines will be documented in the DSMB charter.

There are no formal statistical stopping rules, however the DSMB will have the responsibility for independently evaluating safety on the bases of there being no evidence of safety concern(s) to warrant study cessation. The occurrence of bone marrow failure (defined as a protracted neutropenia (ANC < 0.5x10<sup>3</sup>/µL (mm<sup>3</sup>)) and/or thrombocytopenia (platelets < 25x10<sup>3</sup>/µL (mm<sup>3</sup>)) after Week 12 post-infusion) will trigger a temporary hold on the administration of busulfan and subject enrolment pending a safety assessment by the DSMB. The occurrence of grade 4 laboratory abnormalities, unanticipated incidence, severity or frequency of AE/SAEs, or failure of Ttn/HSPCtn manufacturing processes may also be events that could present sufficient safety concerns to warrant study cessation. Following completion of the safety data review, the DSMB may also recommend that the study be modified to improve monitoring of safety, additional subjects be enrolled to assess safety, or the study be terminated for safety reasons.


In addition to scheduled review of Cohort data, the DSMB chairperson will receive a copy of all MRC recommendations and all SAE reports that have possible suspect causality to Cal-1 and/or the study procedures in real time (i.e. at the same time as the MRC). The Chairperson is responsible for determining if a special meeting of the DSMB is required to review any event in further detail and make a recommendation between cohorts. Recommendations will be submitted to the Sponsor and authorities as required, according to local guidelines and regulations.

There are two planned DSMB safety analyses and one preliminary analysis for safety and secondary endpoints at Week 24. The independent DSMB will conduct a complete review of data to Week 12 for at least 3 subjects in the preceding Cohort before subjects in Cohorts 2 and 3 receive any busulfan and are infused. At each analysis, all subjects' safety data will be summarized including all available data up to the time the analysis is conducted. Measures of Cal-1 marking/expression will also be summarized. There will be no formal statistical stopping rules, rather the study will continue on the basis of there being no evidence of sufficient safety concerns to warrant study cessation. The occurrence of bone marrow failure (defined as a protracted neutropenia (ANC < 0.5x10<sup>3</sup>/µL (mm<sup>3</sup>)) and/or thrombocytopenia (platelets <  $25x10^3/\mu L$  (mm<sup>3</sup>)) after Week 12 post-infusion), the occurrence of grade 4 laboratory abnormalities, unanticipated incidence, severity or frequency of AE/SAEs, or failure of T<sup>tn</sup>/HSPC<sup>tn</sup> manufacturing processes may be events that could present sufficient safety concerns to warrant study cessation. Efficacy indicators, such as the degree of Cal-1 marking in peripheral blood, GALT and bone marrow will also be assessed.

# 16.3.Interim Analyses

A formal preliminary analysis was planned to be conducted once all subjects completed 24 weeks follow-up. No formal preliminary analysis was conducted by CC Calimmune's request. Safety and efficacy data review was conducted by the MRC for all subjects who completed 24 weeks follow up and beyond.

### 16.4. Final Analysis (End of Study).

Formal final analyses will be performed at the end of the study generating Statistical Analysis System (SAS) tables, figures and listings for use in drafting the CSR as described in the SAP. These will be considered the final analyses.

The final end of study analysis (i.e. results post lock of the data base) will be based on the final version of the SAP.


# 17.Software

The following software will be used to perform the statistical analyses: SAS® Version 9.4 or higher (SAS Institute, Cary, North Carolina, USA).


# 18.Tables

| No. | Title | Analysis<br>Population |
|---|---|---|
| 1 | Protocol Deviations | All Enrolled |
| 2.1 | Protocol Deviations: Major Deviations Summary | All Enrolled |
| 2.2 | Protocol Deviations: Minor Deviations Summary | All Enrolled |
| 3 | Demographic and Baseline Information | All Enrolled |
| 4 | HIV-1 History | All Enrolled |
| 5 | Manufacturing CD4+ – Cohorts 1 and 2 and 3 | Safety |
| 6 | Manufacturing CD34+ – Cohorts 1 and 2 and 3 | Safety |
| 7 | Manufacturing Deviations | Safety |
| 8 | Cell Dose (x10e8) at Day 0 vs. Marking/Expression Data | Safety |
| 9 | Busulfan AUC (uMol/min) vs. Marking/Expression Data | Safety |
| 10.1 | CD4+ Count (mm <sup>3</sup> ) | Safety |
| 10.2 | CD4+ Count mm³) vs. Marking/Expression Data | Safety |
| 10.3.1 | HIV-1-RNA Roche Assay (copies/mL) | Safety |
| 10.3.2 | HIV-1-RNA Abbott Assay (copies/mL) | Safety |
| 10.4.1 | HIV-1-RNA Roche Assay (copies/mL) vs. Peak<br>Marking/Expression Data | Safety |
| 10.4.2 | HIV-1-RNA Abbot Assay (copies/mL) vs. Peak Marking/Expression Data | Safety |
| 11.1 | ANC (10 <sup>3</sup> /uL) vs. Peak Marking/Expression Data | Safety |
| 11.2 | Platelets (10 <sup>3</sup> /uL) vs. Peak Marking/Expression Data | Safety |
| 12 | Lymphocyte Development and Chronic Inflammation vs. Marking/Expression | Safety |
| 13.1 | Adverse Events (Summary SOC, PT) | Safety |
| 13.2 | Adverse Events by CTC grade (Severity) | Safety |
| 13.3 | Treatment Emergent Adverse Events by Relationship to Study Drug (Causality) | Safety |
| 13.4 | Adverse Events by Relationship to Study Procedure (Causality) | Safety |


# 19.Listings

| No. | Title | Analysis<br>Population |
|---|---|---|
| 1 | Subject Disposition | All Enrolled |
| 2 | Subject Withdrawal | All Enrolled |
| 3 | Subject Discontinuation | All Enrolled |
| 4.1 | Demographics | All Enrolled |
| 4.2 | Pre-Busulfan Body Weight | All Enrolled |
| 5 | HIV-1 History | All Enrolled |
| 6 | Medical History | All Enrolled |
| 7 | Eligibility Criteria | All Enrolled |
| 8.1 | Pregnancy Test | All Enrolled |
| 8.2 | Positive Pregnancy Test | All Enrolled |
| 9 | Chest X-Rays | All Enrolled |
| 10 | ART Therapy History (regimen overview) | All Enrolled |
| | Transduced CD4+ Cell Product Dose (Transduction | All Enrolled |
| 11 | efficiency, viability, cell numbers for Ttn) | |
| 12 | Transduced CD34+ Cell Product Dose (Transduction efficiency, viability, cell numbers for HSPC <sup>tn</sup> ) | All Enrolled |
| 13.1 | Plerixafor Therapy | All Enrolled |
| 13.2 | G-CSF Therapy | All Enrolled |
| 14.1 | Apheresis – CD4+ | All Enrolled |
| 14.2 | Apheresis – CD34+ | All Enrolled |
| 15.1 | Busulfan Dosing | |
| 15.2 | Busulfan Administration and Pharmacokinetics | All Enrolled |
| 16 | Cal-1 Marking/Expression - Peripheral Blood | All Enrolled |
| 17 | Cal-1 Marking/Expression - Bone Marrow | All Enrolled |
| 18 | Cal-1 Marking/Expression – GALT | All Enrolled |
| 19.1 | Cal-1 Marking/Expression – Subsets: Monocytes | All Enrolled |
| 19.2 | Cal-1 Marking/Expression – Subsets: Granulocytes | All Enrolled |
| 19.3 | Cal-1 Marking/Expression – Subsets: CD4+ Lymphocytes | All Enrolled |
| 19.4 | Cal-1 Marking/Expression – Subsets: CD8+ Lymphocytes | All Enrolled |
| 20.1 | Serious Adverse Events, including event narratives | All Enrolled |
| 20.2 | Deaths | All Enrolled |
| 21.1 | Adverse Events (All Grades) | All Enrolled |
| 21.2 | Adverse Events (Grades 3 and /or 4) | All Enrolled |
| 21.3 | Related Adverse Events (Grades 3 and /or 4) | All Enrolled |
| 22.1 | Concomitant Medication | All Enrolled |
| 22.2 | Concomitant Procedures and Therapies | All Enrolled |
| 23.1 | Laboratory – Hematology | All Enrolled |
| 23.2 | Laboratory – Hematology (Abnormal only) | All Enrolled |
| 24.1 | Laboratory – Biochemistry | All Enrolled |
| 24.2 | Laboratory – Biochemistry (Abnormal only) | All Enrolled |
| 25.1 | Laboratory – Lymphocyte phenotype | All Enrolled |
| 25.2 | Laboratory – Thymopoieisis | All Enrolled |
| 25.3 | Laboratory – Inflammation | All Enrolled |
| 25.4 | Laboratory – Maturation | All Enrolled |
| 26 | Laboratory – HIV-1 RNA | All Enrolled |
| 27.1 | Vital Signs | All Enrolled |


| No. | Title | Analysis<br>Population |
|------|----------------------------------------|------------------------|
| 27.2 | Abnormal Vital Signs | All Enrolled |
| 28.1 | Physical Examination | All Enrolled |
| 28.2 | Abnormal Physical Examination | All Enrolled |
| 29.1 | Cal-1 Integration Analysis | All Enrolled |
| 29.2 | Cal-1 Integration Analysis (Re-test) | All Enrolled |
| 30 | Replication Competent Lentivirus (RCL) | All Enrolled |
| 31 | HIV-1 Tropism Assay | All Enrolled |
| 32.1 | C46 Immunogenicity – Humoral Response | All Enrolled |
| 32.2 | C46 Immunogenicity – Cellular Response | All Enrolled |

Protocol Number: CAL-USA-11 Document status: Final SAP Version 1.0

# 20.Figures

| No. | Title | Analysis<br>Population |
|---|---|---|
| 1.1.1 | T <sup>tn</sup> (CD4+) Cell Dose at Day 0 vs. Peak Marking/Expression Data Protocol: CAL-USA-11 | Safety |
| 1.1.2 | T <sup>tn</sup> (CD4+) Cell Dose at Day 0 vs. Week 48 Marking/Expression Data | Safety |
| 1.2.1 | HSPC <sup>tn</sup> (CD34+) Cell Dose at Day 0 vs. Peak<br>Marking/Expression Data | Safety |
| 1.2.2 | HSPC <sup>tn</sup> (CD34+) Cell Dose at Day 0 vs. Week 48 Marking/Expression Data | Safety |
| 2.1.1 | Busulfan AUC (uMol/min) at Day -4 vs. Peak Marking/Expression | Safety |
| 2.1.2 | Busulfan AUC (uMol/min) at Day -4 vs. Week 48 Marking/Expression Data | Safety |
| 2.2.1 | Busulfan AUC (uMol/min) at Day -2 vs. Peak Marking/Expression | Safety |
| 2.2.2 | Busulfan AUC (uMol/min) at Day -2 vs. Week 48 Marking/Expression Data | Safety |
| 3.1.1 | CD4+ Count (mm³) at Screening vs. Peak Marking/Expression Data | Safety |
| 3.1.2 | CD4+ Count (mm3) at pre-Apheresis vs. Peak Marking/Expression Data | Safety |
| 3.1.3 | CD4+ Count (mm³) at pre-infusion (Cohort 1) /pre-busulfan (Cohorts 2 and 3) vs. Peak Marking/Expression Data | Safety |
| 3.1.4 | Peak CD4+ Count (mm³) change from Screening vs. Peak Marking/Expression Data | Safety |
| 3.1.5 | Peak CD4+ Count (mm³) change from pre-Apheresis vs. Peak Marking/Expression Data | Safety |
| 3.1.6 | Peak CD4+ Count (mm³) change from pre-infusion (Cohort 1) /pre-busulfan (Cohorts 2 and 3) vs. Peak Marking/Expression Data | Safety |
| 3.1.7 | Week 48 CD4+ Count (mm³) change from Screening vs. Peak Marking/Expression Data | Safety |
| 3.1.8 | Week 48 CD4+ Count (mm³) change from pre-Apheresis vs. Peak Marking/Expression Data | Safety |
| 3.1.9 | Week 48 CD4+ Count (mm³) change from pre-infusion (Cohort 1) /pre-busulfan (Cohorts 2 and 3) vs. Peak Marking/Expression Data | Safety |
| 3.2.1 – 3.2.9 | As per 3.1.1 – 3.1.9 for Week 48 Marking/Expression Data | Safety |
| 3.3.1 – 3.3.9 | As per 3.1.1 – 3.1.9 for HIV-1-RNA (copies/mL) vs. Peak Marking/Expression Data | Safety |
| 3.4.1 – 3.4.9 | As per 3.1.1 – 3.1.9 for HIV-1-RNA (copies/mL) vs. Week 48 Marking/Expression Data | Safety |
| 4.1.1 – 4.1.9 | As per 3.1.1 – 3.1.9 for nadir ANC (10³/uL) vs. Peak Marking/Expression Data | Safety |
| 4.2.1 – 4.2.9 | As per 3.1.1 – 3.1.9 for nadir ANC (10³/uL) vs. Week 48 Marking/Expression Data | Safety |
| 4.3.1 – 4.3.9 | As per 3.1.1 – 3.1.9 for Platelets (10³/uL) vs. Peak Marking/Expression Data | Safety |


| No. | Title | Analysis<br>Population |
|---|---|---|
| 4.4.1 – 4.4.9 | As per 3.1.1 – 3.1.9 for Platelets (10 <sup>3</sup> /uL) vs. Week 48 Marking/Expression Data | Safety |
| 5.1.1 – 5.1.9 | As per 3.1.1 – 3.1.9 for Lymphocyte Development and Chronic Inflammation vs. Peak Marking/Expression Data | Safety |
| 5.2.1 – 5.2.9 | As per 3.1.1 – 3.1.9 for Lymphocyte Development and Chronic Inflammation vs. Week 48 Marking/Expression Data | Safety |
| 6 | Busulfan Pharmacokinetics, AUC and Clearance Rate | Safety |
| 7.1 | Post busulfan – WBC (10³/uL) | Safety |
| 7.2 | Post busulfan – ANC (10 <sup>3</sup> /uL) | Safety |
| 7.3 | Post busulfan – Platelets (10³/uL) | Safety |
| 8.1 – 8.2 | %CD3/CD4 by Cohort | Safety |
| 8.3 - 8.4 | %CD3/CD8 by Cohort | Safety |
| 8.5 - 8.6 | Absolute CD3/CD4 by Cohort | Safety |
| 8.7 - 8.8 | Absolute CD3/CD8 by Cohort | Safety |
| 8.9 – 8.10 | CD4:CD8 Ratio by Cohort | Safety |
| 9.1 – 9.8 | HIV-1 RNA (copies/mL) by Subject | Safety |
| 9.9 - 9.10 | HIV-1 RNA (copies/mL) Roche log <sub>10</sub> by Cohort | Safety |
| 10.1 – 10.2 | Peripheral Blood Marking by Cohort | Safety |
| 10.3 – 10.4 | CD4 Marking by Cohort | Safety |
| 10.5 – 10.6 | CD8 Marking by Cohort | Safety |
| 10.7 – 10.8 | Granulocytes by Cohort | Safety |
| 10.9 – 10.10 | Monocytes Marking by Cohort | Safety |
| 10.11 – 10.12 | Bone Marrow Marking by Cohort | Safety |
| 10.13 – 10.14 | GALT Marking (Location 1) by Cohort | Safety |
| 10.15 – 10.16 | GALT Marking (Location 2) by Cohort | Safety |
| 11 | Kaplan Meier Plot of Time to ART start | Safety |


# 21.References

1. Clinical Study Protocol Version 8, dated 08 JUL 2015.
Protocol Number: CAL-USA-11 Document status: Final SAP Version 1.0

## 22. Appendix I: Summary of Protocol Changes

CAL-USA-11 PROTOCOL VERSION 3.0 (dated 12 December 2013) - SUMMARY OF CHANGES

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Contact information | Update | |
| Glossary of terms | Update/addition | New terms added. Changed SUA to SUSAR. |
| Synopsis | Addition | Added clinical trials.gov registration number Added participating countries (USA). |
| | Update | All units for laboratory values were updated to ISO (conventional) format for consistency. |
| Schedule of Events | Modification & addition | <ul> <li>Separated tables to pre-infusion and post-infusion</li> <li>Pre-infusion:</li> <li>1. Added option pre-screening to help facilitate selection of suitable potential subjects and reduce the screenfail rate</li> <li>2. Separated consent procedure to ensure consent obtained prior to pre-screening</li> <li>3. Increased window period for Screening 1 visit to assist sites in the consenting and scheduling of concurrent subjects for screening</li> <li>4. Moved co-infection screening to Screening 1 due to better accommodate assay turn-around times and the Screening 2 window period</li> <li>5. Added busulfan PK monitoring in response to FDA and DSMB request</li> <li>6. Increased the window between CD34 apheresis and Baseline visit to better accommodate the turn-around time for product release testing</li> <li>Post-infusion:</li> <li>1. Added 'Conditioning F/U' visits at week 0.5, 1.5, 2.5, 3, 3.5, 4.5, 5, and 5.5 time points to increase intensity of post-conditioning and transplant subject safety monitoring in response to FDA request and in line with DSMB recommendations</li> <li>Footnotes:</li> <li>1. Updated in line with above changes and change to lymphocyte phenotyping studies (see section 7.5).</li> <li>2. Added unscheduled HIV-1 tropism assessment if subject discontinues the study post-infusion to recommence ART (see section 6.2.4)</li> <li>3. Added stored EDTA-plasma sample for HIV viral load batch analysis (see section 7.5).</li> </ul> |

Protocol Number: CAL-USA-11

| Protocol Section | Nature of Change | Rationale |
|---|---|---|
| 1.1 Background | Addition | In vivo studies added to section 1.1.1. Additional references cited section 1.1.2 literature update. Additional references cited section 1.1.2 (busulfan) regarding the use of low and intermediate doses of busulfan for non-myeloablative and reduced-intensity conditioning effects. |
| 3. Objectives and Outcome measures/endpoints | Modification | Update in line with changes to lymphocyte phenotyping studies (per section 7.3). |
| 4.Overview of study design | Modification | Updated timeline schematic in line with changes to the pre-infusion schedule of events. Updated DSMB recommendations to include Cohort 3 proceeding with an increased dose of 6 to 8mg/kg busulfan (See section 6.2.2) |
| 5.2 Exclusion criteria | Modification | Ex-A updated to be in ISO units Ex-N modified to specify venous assessment <u>prior</u> to Screening1, to allow flexibility in scheduling. |
| 5.4 Rescreening | Modification | Re-screening procedures were adjusted in line with the changes to Screening 1 and Screening 2 procedures. |
| 6.1.3 Dosage and administration | Modification | The order of infusion was changed to administer the HSPC <sup>tn</sup> first. This was a safety consideration, as an adverse reaction to the infusion products is potentially more likely with the T <sup>tn</sup> . HSPC <sup>tn</sup> are the priority infusion for subjects who have received busulfan conditioning. The order of infusion for Cohort 1 subjects was T <sup>tn</sup> , followed by HSPC <sup>tn</sup> . |

| Protocol Section | Nature of Change | Rationale |
|---|---|---|
| 6.2.2 Busulfan | Modification | The dosing range for busulfan was modified to include 6mg/kg within the 'moderate dose' cohort (III). Dose adjustment rules, based on observation of delayed hematopoietic recovery were added. These changes are an additional safety precaution to ensure the dose of busulfan does not result in a more severe myeloablation than intended. The description of the busulfan dosing was corresponding updated throughout the protocol. As a safety precaution to ensure there would be sufficient CD34+ cells to 'rescue' a subject in the event of busulfan-induced myeloablation, a clause was added that busulfan will not be administered if the minimum anticipated HSPC <sup>tn</sup> dose (0.5x10 <sup>8</sup> total CD34+ cells) is not achieved. If cell infusion is postponed, the administration of busulfan will also be postponed. Busulfan will be given 2 days prior to the revised planned cell infusion date (baseline visit) with the contingent that all release criteria were met. |
| 6.2.3 Post-busulfan infection prophylaxis | Addition | New section added to include specification on the post-<br>conditioning infection prophylaxis regimen. Details of<br>agents, doses and duration are provided. |
| 6.2.4<br>Antiretroviral Therapy | Addition | HIV-1 tropism will also be performed if a subject is required to recommence ART post-infusion. |
| 7.1.1 Consent | Addition | New section created to align with the re-design of the schedule of events. Details are provided on the permitted timing of study consent. |
| 7.1.2 Pre-screening | Addition | New section created to align with the re-design of the schedule of events. The pre-screening visit is an optional visit included to assist sites in the selection of potential suitable subjects to participate. Consent requirements, optional visit procedures/laboratory tests and timing are described. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 7.1.3 Screening 1 | Modification | A screen fail rate of > 50% was experienced with Cohort 1. Screen failures present a risk and inconvenience to study subjects and also increase study timelines. The timing of Screening has been adjusted to allow a maximum 3 month interval between consent and Screening 1 (increase from 2 months) to allow sites more time to obtain and evaluate pre-existing medical history as part of eligibility and suitability determination. Procedures were revised to include the co-infection screening and chest x-ray (moved from Screening 2). This was to simplify the screening 2 procedures, to minimise the risk of late notice screen fails and therefore reduce impact on both the individual subjects and the manufacturing facility preparation. A window period was added for the venous assessment, to allow this to be performed any time between consent and Screening 1. This will improve subject convenience, and also enable assessment of this eligibility criterion before the more invasive assessments are performed. Medical history instructions were expanded to specify collection of vaccination, drug allergy and recurrent infection history, in line with standard bone marrow transplant procedures |
| 7.1.4<br>Screening 2 | Modification | Window period modified to be within 1-2 weeks of CD4 apheresis. Window between Screening 1 and Screening 2 modified to 2-12 weeks to allow concurrent screening (within limitations specified in Section 12.1). Visit laboratory tests simplified to confirmation of HIV-1 RNA and CD4+ eligibility criteria. Chest x-ray and coinfection screening moved to Screening 1 because of assay turn-around times. |
| 7.1.5<br>CD4+ T lymphocyte<br>apheresis | Modification & addition | Added subject's weight to be measured and provided to the manufacturing lab to enable calculation of the anticipated dose for the finished T <sup>tn</sup> product. CCI Removed description of tests to be performed on the collected apheresis product, as these are manufacturing-specific procedures. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 7.1.7<br>CD34 + apheresis | Modification & addition | Added subject's weight to be measured and provided to the manufacturing lab to enable calculation of the anticipated dose for the finished HSPC <sup>tn</sup> product |
| | | Removed description of tests to be performed on the collected apheresis product, as these are manufacturing-specific procedures. |
| 7.1.8<br>Administration of<br>busulfan | Modification & addition | Added stipulation that this visit can only occur after confirmation that the T <sup>tn</sup> and HSPC <sup>tn</sup> products have been released and are available on site |
| | | Clarified the timing of each busulfan dose to be in the morning |
| | | Added instruction in the event of a delay in the planned cell infusion (Baseline) visit |
| | | Added specification for collection of blood samples and batch testing for busulfan PK monitoring. |
| 7.1.9<br>Baseline (day of<br>infusion) | Modification | Removed the provision to postpone the infusion if busulfan conditioning has occurred |
| | | CCI |
| 7.2.1<br>Conditioning follow<br>up | Addition | New section to describe the content and timing of additional visits to increase intensity of post-conditioning and cell-infusion safety monitoring. Both laboratory and clinical monitoring is specified Extended or more frequent safety follow up is permitted if clinically indicated for any study subject. |
| 7.2.2 Weeks 1, 2, 6, 8,<br>16 & 20 | Addition | Provision to perform a local STAT CBC/differential has been added to Weeks 1, 2 and 6, in line with conditioning follow up visits in section 7.2.1 Safety limits are provided, along with appropriate steps to ensure subjects are further evaluated and – as necessary – treated by an experienced, accredited transplant center. |
| 7.2.3 Week 4 | Addition | Provision to perform a local STAT CBC/differential has been added, in line with conditioning follow up visits in section 7.2.1 |

| Protocol Section | Nature of Change | Rationale |
|---|---|---|
| 7.3 Safety evaluations | Modification & addition | C46 immunogenicity studies were moved from exploratory analysis (Section 7.6) to safety, in line with FDA request to perform these studies as part of the Cal-1 safety data collection. |
| 7.5<br>Efficacy evaluations | Modification & addition | Lymphocyte phenotyping studies have been added and grouped under the heading of 'Lymphocyte development studies'. In addition to the thymopoiesis analysis, these now include 'maturation' and 'inflammation' to expand potential data on the impact of Cal-1 on lymphocyte dynamics. An additional baseline time point at the CD4+ apheresis visit was added to obtain baseline prior to apheresis and G-CSF mobilization. Potential cross-reactivity with Cal-1 in HIV-1 viral load assays has been identified as an area for further laboratory investigation. The HIV-1 RNA plasma assay details have been updated with the addition of a stored EDTA-plasma sample for the purposes of batch analysis with an alternative FDA approved plasma HIV-1 RNA assay, pending the outcome of these investigations. Corresponding updates to the Schedule of Events, visit-specific procedures and statistical analysis have been made for consistency throughout the protocol. |
| 7.6<br>Exploratory<br>evaluations | Modification & addition | |
| 7.7 Specimen storage | Modification | Storage of blood and tissue samples was previously described within the exploratory evaluations section. This has been moved into a separate section for clarity. Priority of use of the stored specimens has been clarified. |
| 10.1.4 | Modification | The term Serious Unexpected Associated (SUA) Adverse Event was replaced with Serious & Unexpected Suspected Adverse Reaction (SUSAR) to be consistent with regulatory guidance and other study-related safety operational documentation (such as the DSMB charter and safety management plan) The term SUSAR replaces SUA throughout the protocol for consistency. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 11.2<br>Ethical and regulatory<br>information | Addition | Details of the IND # and clinicaltrials.gov registration were added DSMB recommendation was added to the list of informational study updates to be provided to investigators. |
| 11.5<br>Privacy and<br>confidentiality | Addition | Reference to adherence to HIPPA regulations was added. |
| 12.1<br>Subject screening and<br>enrolment | Addition | Provision has been added to allow the concurrent screening of subjects in order to minimize the potential negative impact of screen failures on the participating subjects, sites and manufacturing schedules. The total number of subjects in screening at any time cannot exceed the number of available places within the cohort. Details on the timing and scheduling of subject visits is addressed. |
| | | Consequent changes to the schedule of events and visit specific information are addressed throughout the protocol for consistency. |
| 12.7.1 MRC | Addition | Specification was added for the MRC review of hematopoietic recovery post busulfan and for the MRC to document their recommendation concerning an adjustment of the busulfan dose within the range specified. |
| 12.7.2 DSMB | Addition | Bone marrow failure has been defined by hematologic parameters and added as a stopping rule in addition to the events previously listed. Provision is also added for the DSMB chairperson to receive copies of MRC recommendations in real-time, and scope added to convene a special meeting of the DSMB and recommendations to be made between formal cohort reviews. |
| 12.10.1<br>Sources of funding<br>and disclosure of<br>financial interest | Modification | Section updated to include information on source of Calimmune financial support, including disclosure of a CIRM grant. |
| Appendix I | Modification | In order ensure up to date information, the DAIDS grading tables have been deleted and replaced with a link to the on line published document. The current version is December 2004, with clarifications dated August 2009. Specific guidance for values below Grade 1 have been added, in line with the DAIDS instructions. |

| Protocol Section | Nature of Change | Rationale |
|---|---|---|
| Appendix III | Modification & addition | |
| Appendix IV | Modification | <ul> <li>Section 3</li> <li>updated with details on prophylactic medications, dose and timing</li> <li>flow rate reduced to deliver total dose over 4 hours</li> <li>Section 5 updated with medications list.</li> </ul> |
| Appendix V | Modification & addition | Specific apheresis collection parameters provided for both CD4+ and CD34+ collections. |

Protocol Number: CAL-USA-11 15 December 2017

CAL-USA-11 PROTOCOL VERSION 4.0 (dated 22 March 2014) – SUMMARY OF CHANGES

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Schedule of events | Removed<br>footnotes referring<br>to 4-week acute<br>and 12-week sub-<br>acute data time<br>points | Original footnotes were potentially misleading. It is intended that data inclusive to Week 12 (not only weeks 4 and 12) to be presented to the DSMB. |
| | Busulfan PK<br>monitoring<br>footnote revised | Details on PK sampling now described in Appendix IV. Additionally, it was clarified that for Cohort 3, the busulfan dosing will start on Day -3 (and therefore completing at the same time relative to infusion as Cohort 1). Corresponding updates to text made throughout the document to correct references to Day -2 and Day-3 |
| | Additional column<br>for busulfan (Day -<br>3) | Additional column added to separate the 2 days of busulfan and highlight the difference between cohorts 2 and 3 |
| | Footnote 18<br>(unscheduled HIV-<br>1 tropism) deleted | Unscheduled HIV-1 tropism no longer to be performed.<br>Footnote 19 (Plasma HIV-1 RNA) renumbered to 18 |
| | Additional visits:<br>Week 28, 36 & 44 | Additional visits in the final 12 weeks of the follow up period have been added so the frequency of follow up remains 4-weekly. The rationale for this change is that ongoing monthly follow up intervals allows closer follow up of HIV-1 viral load and CD4+ T-cell counts. |
| 3. Objectives &<br>Outcome<br>measure/Endpoints | Secondary efficacy<br>data description<br>modified | Format change to better describe evaluation of lymphocyte inflammation studies (separate bullet point from thymopoiesis and maturation). Various text updates then required throughout for consistency. |
| 4.1 Overview | Minimum number of subjects per cohort reduced from 4 to 3. DSMB review consequently will proceed on data from 3 subjects, with an option for a fourth subject if requested. | There has been a higher than expected screen failure rate (70%) and correspondingly an overall delay in study timelines. The original subject numbers were not based on formal power considerations, and no major safety concerns have presented to date. Thus, the change in sample size is being made in order to restore study timelines, yet not significantly impacting the probability of obtaining meaningful safety data from the study. Various text updates then required throughout for consistency. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 5.1 General<br>Considerations | Timing for commencement of each subsequent cohort revised | Screening for the next cohort will not commence until after the data for 3 subjects to Week 12 of post-infusion follow up is available for the DSMB review. |
| 6.2.2 Busulfan / 12.7.1<br>MRC / 12.7.2 DSMB | Text changes for consistency. | Busulfan dose adjustment and temporary hold on further dosing had been included in the protocol with version 3.0 changes. There were however small inconsistencies between the relevant sections that have now been addressed, and both dose adjustment or a hold on dosing are possible options for the MRC and DSMB in the event delayed hematopoietic recovery or/and bone marrow failure is observed with any subject. |
| 6.2.4 Antiretroviral<br>Therapy | Specific instructions added with respect to the confirmatory retest in the event that s subjects HIV-1 viral load exceeds the specified safety limit. | Cross-reactivity with the Cal-1 vector has been demonstrated in the Roche COBAS® AmpliPrep/COBAS® TaqMan® HIV-1 RNA PCR assay. Because this cross-reactivity has the potential to artificially elevate viral load results, the confirmatory assay is to be performed with an alternative HIV-1 assay (Abbott RealTime m2000), which does not appear to cross-react with the Cal-1 vector. To ensure accurate interpretation of results, complete batch analysis of all time points is specified in the event a confirmatory re-test is required. Abbott RealTime m2000 batch data will be used for formal analyses. |
| 7.1.8 Administration of Busulfan | Details of PK sampling removed | Details on sampling have been removed from this section and now described in Appendix IV. |
| 7.3 Safety Evaluations | Reference to RCL<br>biological assay<br>removed | As both Cal-1 vector and the disease indication are a lentivirus, biological RCL assay is not technically feasible. |
| 7.5 Efficacy<br>Evaluations | Details of cross-<br>reactivity updated,<br>with specific<br>alternative assay<br>added<br>Further details on<br>Cal-1 marking | Cross reactivity with Cal-1 has been confirmed and the Abbott RealTime m2000 assay has been identified as a suitable alternate assay for batch analysis. Clarified the PCR targets for monitoring of Cal-1 presence and activity |
| | Cal-1 marking<br>&expression added | and activity |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 8. Subject Withdrawal/Discontin uation | Definition of discontinuation and withdrawal clarified | Discontinuation has been clarified as referring to the population of subjects that are discontinued from secondary analysis due to commencement of ART or other prohibited concomitant medication. These subjects continue in safety follow up. Withdrawal has been clarified as referring to the population of subjects that have ceased study participation. Various text updates then required throughout for consistency, particularly section 9.1. |
| 9. Statistical Methods | Power calculations updated with new subject numbers | Changes to text within the Safety and Key Efficacy sections made to include power calculations for 3 subjects per cohort as well as 4 |
| 9.1 Statistical Analysis | Clarification on<br>which assay data<br>to be used in<br>formal analyses | Formal statistical analysis will be performed using the batch data from the Abbott assay. |
| 12.7.2 DSMB | Clarification added<br>regarding data for<br>DSMB review and<br>scope of<br>recommendations | Removed reference to acute and sub-acute time points (per Schedule of Events), and revised section text accordingly. Added description of the potential scope for DSMB recommendation to include improved safety monitoring, study modification, additional subject recruitment and termination. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Appendix IV | PK sampling information added | PK sampling moved from section 7.1.8 to include together with other instructions on the administration and monitoring of busulfan. The PK sampling schedule was improved with additional collection time points. Additionally, the site for PK blood draw details were expanded to increase consistency across sites in collection and handling of samples. For logistical reasons, a window period of 3 days prior to Day -2 has been added for subject's weight for the purposes of busulfan dose calculation. |
| | Other significant changes made to improve safety and enhance clarity for implementation | <ul> <li>Changes to the busulfan preparation, administration and monitoring include: <ul> <li>Adjusted ideal body weight dose calculation, and specification on value to use for dose calculation.</li> <li>Further specifications provided to provide clarity for pharmacists and clinical staff (e.g. use of an IV tube filter, infusion timing, IV placement etc.).</li> <li>For operator safety, the IV line is to be primed with saline (not busulfan), and an over-fill has been added to the infusion volume to adjust for the IV line volume.</li> <li>Needle size and infusion time reduced in line with standard practice.</li> <li>Lorazepam replaced with levetiracetam (Keppra™) as the prophylactic agent for busulfaninduced seizure. Levetiracetam is less sedating and provides safe and stable seizure prophylaxis.</li> <li>Extended anti-emetic medication to include PRN oral dosing in addition to IV pre-medication.</li> <li>Timing of vital signs adjusted to make more consistent though the total infusion and PK period.</li> <li>Specified additional prohibited concomitant medications that may interfere with busulfan clearance.</li> </ul> </li> </ul> |

CAL-USA-11 PROTOCOL VERSION 5.0 (dated 12 June 2014) – SUMMARY OF CHANGES

| Protocol Section | Nature of Change | Rationale |
|---|---|---|
| Protocol Section Section 6.1.1 Section 6.1.3 Appendix III | Nature of Change Update anticipated dose of T <sup>tn</sup> (cell numbers and volume) | Rationale |
| Section 6.1.1.2<br>Section 6.2.2<br>Section 7.1.8<br>Section 7.1.9<br>Appendix III | CD34 minimum<br>dose revised | Previously expressed as a total number of cells, the minimum dose of HSPC required to proceed with busulfan conditioning has been revised to be expressed as a dose per kg of subject weight. An aliquot of 1x106 CD34+ cells/kg will be cryopreserved prior to <i>in vitro</i> manipulations with the manufacture of the HSPCtn dose. These reserved cells will be administered of the HSPCtn dose is less than 2x106/kg. |
| Section 7.1.4 | Updated description of timing between Screening 1 and 2 | Inconsistency between protocol text and SOE addressed by updating section 7.1.4 wording |
| Section 7.1.8 Appendix III Appendix IV | O2 saturation included in busulfan infusion observations | Vital sign monitoring to include O2 saturation during the actual infusions, but not required during the PK collection period. Subjects to continue to be visually monitored during this period, with vital signs to be measured as clinically indicated. |
| Section 7.2.4 Section 8 Schedule of Events Appendix V | Addition of a pre-<br>busulfan<br>assessment visit | A scheduled study visit allows for more comprehensive safety assessment prior to commencement of busulfan |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Section 7.5 | Update description of batch analysis using the Abbott HIV viral load assay | Inconsistency between protocol text and SOE footnotes addressed by updating section 7.5 wording |
| Section 8<br>Schedule of<br>Events | Addition of withdrawal/discontinuation visit | A withdrawal/discontinuation visit allows timely capture of important safety and efficacy data at the time of subject withdrawal/discontinuation visit. |
| Appendix IV | Updated list of contraindicated medications Removed specification for IV size for PK sampling | Azithromycin added to the list of contraindicated medications as it may significantly slow busulfan clearance. Specification for a 22 gauge IV for the PK sampling has been removed, allowing the site discretionary choice of the IV size |

CAL-USA-11 PROTOCOL VERSION 6.0 (dated 14 October 2014) - SUMMARY OF CHANGES

| Protocol | Nature of Change | Rationale |
|---|---|---|
| SOE<br>5.4/5.5<br>6.1.2<br>7.1.5<br>8 | Permit repeat of small volume apheresis in event that the initial T <sup>tn</sup> manufacturing is not successful or some other event prevents release or infusion of the product. | Multiple, small volume aphereses are performed in clinical practice following sufficient time for PBMCs to return to preapheresis levels (~ 4weeks). In event of a manufacturing incident, this provision would allow a subject the option to consent to the repeat apheresis and continue in the study. |
| SOE<br>5.3<br>5.4/5.5<br>6.1.2<br>6.2.1<br>7.1.7 | Permit repeat of G-CSF mobilization and large volume apheresis in event that the initial HSPC <sup>tn</sup> manufacturing is not successful or some other event prevents release or infusion of the product | Repeat apheresis procedures are performed in clinical practice following sufficient time for hematopoietic stem cells to return to pre-apheresis levels (~ 4weeks). In event of a manufacturing incident, this provision would allow a subject the option to consent to the repeat procedures and continue in the study. |
| 5.2 | Redefinition of the HIV<br>RNA (viral load) lower<br>and upper limits of<br>eligibility to account for<br>normal variability of the<br>assay | The viral load assay can have a standard variability of 0.2 $\log_{10}$ . Amended inclusion criteria G to specify "Plasma HIV-1 viral RNA $\geq$ 5,000 copies/ml +/0.2 $\log_{10}$ and $\leq$ 100,000 copies/ml +/- 0.2 $\log_{10}$ at Screening 1 and Screening 2 ( $\geq$ 3,200 copies/ml and $\leq$ 160,000 copies/ml)". Improves the screening process without impact on subject characteristics and safety. |
| SoE<br>7.1.4 | Inclusion of chemistry panel in Screen 2 visit | Feedback from apheresis units has been that electrolytes required within at least 2 weeks of planned apheresis to assist with apheresis settings. Inclusion in the study visit (and consequently central lab arrangement) simplifies procedures for the site and subject. In the event that Screening is performed > 2 weeks prior to the planned apheresis, there is now provision for the site to perform local lab CBC/differential with platelets and serum electrolytes. |

| Protocol | Nature of Change | Rationale |
|---|---|---|
| SoE<br>5.2<br>7.1.4<br>7.1.5 | 'Uncoupling' of Screen 2 visit from commencement of apheresis procedures | In practice, there are a number of factors that can impact scheduling for apheresis. The protocol requirement to link Screening to the apheresis visit was often creating stress on the study participants as well on the clinical, apheresis and laboratory facilities involved, because eligibility was not confirmed until all laboratory tests results were reported. By removing the 2-week time stipulation, there is greater flexibility and time for study sites to receive results of labs confirming subjects' eligibility and scheduling of apheresis visit with their apheresis units, thus improving logistics for the sites, without impact on subject safety. The need to have recent CBC and electrolyte data for apheresis settings has been addressed by the inclusion of an additional supplementary ('Pre-apheresis') visit if Screening 2 is performed >2 weeks prior to the planned apheresis. |
| SoE<br>6.2.2<br>7.1.8 | Increased timing of pre-<br>busulfan visit to up to 7<br>days | Improves logistics for the sites and subjects, without impact on subject safety. |
| Appendix IV | Change nausea prophylaxis dose from 16mg IV Ondansetron (Zofran™) to 8mg IV prior to busulfan then, post- busulfan 4mg to 8 mg orally every 8 hours as needed for nausea, not to exceed a total dose of 24 mg in 24 hours. | Maximum ondansetron dose in 24 hour period is 16 mg (stated in the product information). Upon further review of current practice for stem cell transplant procedures, the new dosing schedule has been advised not to exceed 24mg in 24 hours. This dosing schedule has been advised and approved by the Sponsor Medical Review Committee, and allows follow up oral dosing as required, thus potentially improving management of potential nausea secondary to the busulfan. |
| SoE<br>7.2.2 – 7.2.6 | Additional peripheral blood marking and expression studies at Weeks 1, 2 and 6 | Additional time points allow for better monitoring in the early post-transplant period |
| Appendix I - V | Removed provision to update appendix without a formal protocol amendment | This provision has been removed to improve protocol version control. This change was requested by one study site's IBC. |
| Appendix IV | Modified instructions<br>for storage of diluted<br>busulfan for<br>intravenous infusion | Busulfan diluted in saline for infusion has a limited stability period (approximately 12 hours with refrigeration). Instructions modified to recommend refrigerated storage of diluted busulfan to maximize stability. Stability information added for pharmacy and site reference. |

Protocol Number: CAL-USA-11 15 December 2017

| Protocol | Nature of Change | Rationale |
|---|---|---|
| Appendix V | Added provision for use | Short term central venous catheter placement is included as |
| | of central venous | an option for subjects in whom it is clinically indicated to |
| | access for apheresis, if | improve apheresis collection conditions and/or outcome. |
| | clinically indicated | |

Protocol Number: CAL-USA-11


## CAL-USA-11 PROTOCOL VERSION 7.0 (24 March 2015) – SUMMARY OF CHANGES

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Contact<br>Information | Updates | Changes to sponsor and vendor staff and contact details |
| Glossary of<br>Abbreviations | New information | Additional abbreviations added |
| Schedule<br>of Events:<br>Pre-<br>infusion | Changed use of 'Baseline' to 'Day 0' Change to various visit names Changed how window period for Screening 2 expressed Additional new line items, per protocol changes Specimen storage time point added HIV monitoring tests added to pre- busulfan assessment visit | Avoid confusion with analytical baseline reference points, such as Screening. Changes made throughout protocol text for consistency Updated visit names around mobilization and conditioning for consistency and clarity Change for clarity only Line items for plerixafor, and pre-emptive HLA typing added. Specimen storage added to pre-busulfan assessment visit to enable collection of pre-conditioning 'baseline' storage samples Additional CD4+ T lymphocyte panel and HIV-1 RNA in order to gain a more timely pre-conditioning and pre-infusion reference value. |
| Schedule of<br>Events:<br>Post-<br>infusion | Change to various visit names New visit | Updated visit names around post-busulfan monitoring for consistency and clarity and changed how the window period/visit schedule is expressed for clarity only Follow-up Extension added |
| Section 4 | Schematic updated | Schematic of overall study timeline updated to include changes to mobilization and apheresis procedures, as well as addition of the follow up extension. |
| Section 4.2.1 | Change to apheresis rationale | Summary description of yields to date, providing rationale for proposed mobilization and apheresis schedule changes. |
| Section 4.2.3 & 7.2.7 | New section (Follow-Up Extension) | Addition of an 'extension phase' for up to 12 months after Week 48 to allow ongoing monitoring of HIV data after Week 48 in subjects who complete to Week 48 off ART. If a subject had resumed ART prior to week 48, but then again stopped ART prior to Week 48, they would remain eligible to participate in the extension. Various updates to language throughout for consistency and subsequent subsection re-numbered. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Section 5.2 | Wording change to In-E | Re-phrased the term 'viable ART' to 'virologically-effective ART' for clarity. |
| Section 5.3 | Change to Ex-P Wording change to Ex-V | Expanded to include NSAIDS in the contraindicated medications around the period of mobilisation, apheresis. Expanded to include the 6 week period post-busulfan conditioning |
| | Wording change to LX-V | Change reference to 'baseline' to 'cell infusion (day 0)' |
| Section 5.5 | Changes to provisions for repeat procedures | Expanded potential criteria for repeat of apheresis or mobilization/apheresis procedures to include the event that the minimum HSPC <sup>tn</sup> dose (2.0x10 <sup>6</sup> /kg) is not achieved, or failure of storage or shipment conditions (per changes to section 6.1) Simplified and clarified instructions and timing in the event of a process repeat. |
| Section 6.1.1.2<br>&<br>6.1.3 | Increase dose on un- manipulated back-up apheresis product. | The back-up apheresis product is increased from 1x10 <sup>6</sup> CD34+ cells/kg to 1.2x10 <sup>6</sup> CD34+ cells/kg to make allowances for potential losses during the freeze/thaw and administration process. Increasing the cell number is not expected to deplete the final HSPC <sup>tn</sup> dose, as this product is cryopreserved prior to CD34+ selection/purification. |
| | Change HSPC <sup>tn</sup> anticipated dose to a required minimum dose. | Further to experience with 4mg/kg busulfan in Cohort 2, and the degree of hematopoietic impact observed, a minimum dose of 2.0x10 <sup>6</sup> HSPC <sup>tn</sup> /kg has been specified. This is in line with common bone marrow transplant standards, and also enables preservation of the back-up apheresis product for rescue purposes, if required. Various updates throughout for consistency with this change. |
| Section 6.2 & 12.7.1 | Modification to the 'back- up' apheresis product preparation and intention for use. | With the change to specify a minimum 2.0x106/kg HSPC <sup>tn</sup> dose, the back-up apheresis product is now intended to be retained for the treatment of delayed hematopoietic recovery, or bone marrow failure should that occur in any subject. Subjects will be asked at time of initial consent to indicate if they want their back-up apheresis product to be destroyed or donated to Calimmune for research purposes if it is not required (based on recovery status at 12 weeks post-infusion). Various updates throughout and Appendix III for |
| | | Various updates throughout and Appendix III for consistency with this change. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Section 6.3.2 | New section for addition of plerixafor as a mobilizing agent. | Plerixafor can result in up to 2-fold increase in CD34+ cell yields during apheresis; such a boost in CD34+ cell yields will maximise the potential HSPC <sup>tn</sup> dose as well as minimise the possibility of not achieving the minimum target dose. Use of a single dose of plerixafor on Day 4 of G-CSF after the first apheresis and as late as possible in the day to aim for dosing within 16 hours of the next apheresis. Potential short-term gastro-intestinal side-effects will be limited by use of a single dose and managed with anti-diarrhoeal and anti-emetic medications. Various updates throughout for consistency with this change and renumbering of subsequent sections. |
| Section 6.3.3 | Inclusion of provision for HLA typing. Increased busulfan dose range from 6-8mg/kg to 4-8mg/kg given as 2 doses of 2, 3 or 4mg/kg. | Provision is added at the pre-busulfan assessment visit for each site to collect samples for HLA typing according to their standard clinical practice (i.e. testing is to be performed locally and included as a pass-through cost in the study budget). This a safety provision for the unlikely event the autologous back-up product is not effective and allogeneic transplant is required. Increased busulfan dose range gives flexibility to either continue or revert back to the busulfan dose used in Cohort 2. The DSMB will recommend the starting dose. The MRC has the discretion to reduce the dose in response to observation within the cohort. Various changes throughout for consistency |
| Section 6.3.3 | Modification to the definition 'delayed hematopoietic recovery' to extend the time frame from 21 to 42 days post-infusion. Change in platelet limit in definition of delayed hematopoietic recovery and bone marrow failure. | Grade 4 neutropenia and grade 3 or 4 thrombocytopenia has been observed in the first 3 subjects of Cohort 2. The nadir for all 3 has occurred at Day 18 post –infusion. Originally it was anticipated that the nadir would occur approximately 9 days post-infusion. As this nadir is occurring much later than anticipated, the timeline for definition of delayed hematopoietic recovery correspondingly needs adjustment. The platelet limit is increased from 20x10 <sup>3</sup> /μL to 25x10 <sup>3</sup> /μL, in line with the DAIDS grading scale for grade 4 thrombocytopenia. Various changes throughout for consistency |
| Section 6.3.5 | Removed reference to US Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents. | Guidelines have changed, and no longer specify a threshold CD4+ T lymphocyte count for commencement of ART. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Section 7.1.6 & 7.1.7 | Change to 2 x 15L apheresis collections on Days 4 and 5 of G-CSF will be performed instead of the current 1 x 20L apheresis on Day 5. Include provision to collect 100ml autologous plasma on the first day of CD34 apheresis. Additional | Three of the eight CD34+ manufacturing runs to date (Cohorts 1 & 2) have yielded the desired 2x10 <sup>6</sup> HSPC <sup>tn</sup> /kg dose. Multiple smaller volume apheresis collections are often performed clinically and is expected to result in a higher yield of CD34+ cells than the current single collection, which, along with the changes to the mobilization protocol, will improve the feasibility of achieving the required minimum HSPC <sup>tn</sup> dose. The additional plasma is required for overnight storage of the CD34+ cells from the first apheresis. |
| | blood tests during mobilization Added description of optimal apheresis conditions. | Peripheral blood CD34+ counts added on days 3 and 4 of mobilization and additional biochemistry monitoring, including creatinine clearance, for improved efficacy and toxicity monitoring of the new mobilization protocol. Description added to clarify goal with apheresis collections to minimise both red cell and platelet contamination, to assist with manufacturing processes. Various changes throughout and in the Schedule of Events for consistency |
| Section 7.2.1 | Manual<br>differential<br>specified | To improve reliability of local laboratory results, specification for a manual differential added to the required STAT CBC/differential during the busulfan follow up period. |
| Section 7.2.5 | Additional bone<br>marrow and GALT<br>biopsies | Additional biopsies will improve the available data on engraftment and distribution of the transplanted Cal-1-modified cell. Feedback from Investigator's is that the biopsy procedures have been well tolerated. Bone marrow aspirate and GALT biopsies added to Weeks 24 and 48, as well as early discontinuation at the discretion of the Investigator. Various changes throughout, including Schedule of Events and Appendix V for consistency. |
| Appendix II | Update to list of prohibited medication | Clarification around the use of systemic glucocorticisteriods and updates to listed biological immunomodulatory agents and immunostimulants. |
| Appendix IV | Updates to contraindicated medication and delivery specifications | Clarification added around use of common analgesia which is contraindicated with busulfan administration, or during the busulfan recovery period. Removed specific gauge requirement for the IV administration set, allowing investigator discretion. |


Protocol Number: CAL-USA-11

## CAL-USA-11 PROTOCOL VERSION 8.0 (08 July 2015) – SUMMARY OF CHANGES

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Overview of<br>Study Design | Changed description of Cohort 3 dosing to include second dose based on real-time pharmacokinetic-guided dosing to reach targeted drug exposure (AUC). | Recommendation of the DSMB at the June 24, 2015 data review meeting to utilize a targeted busulfan dosing strategy (target of 8000 µMol/L*min based on PK) vs a fixed dose scheme at the 6mg/kg level, as a reduced intensity regimen. |
| Schedule of<br>Events: Pre<br>Infusion | Pre busulfan assessment<br>visit updated to reflect<br>≤11 days | Updated to correct for error in previous protocol version and adjust for change to Day -4 for first dose on busulfan in Cohort 3. Intent remains unchanged to perform pre conditioning assessment within 7 days prior to schedule busulfan infusion. |
| | Changed Cohort 3, 1 <sup>st</sup> dose of busulfan to Day -4 from Day -3 | Allows for needed turn-around-time for real-time PK analysis of 1 <sup>st</sup> day (Day -4) busulfan dose in order to calculate targeted 2 <sup>nd</sup> busulfan dose (Day -2). |
| | Added wording to clarify Day -4 busulfan administration is for Cohort 3 only and Day -2 busulfan dosing for Cohort 2 & 3 | Change for clarity. Updated to correct for errors in previous protocol version. |
| | Updated various superscript footnote numbers Footnote 9 – changed to clarify that at visits G-CSF 3 and G-CSF 4 & plerixafor and CD34 <sup>+</sup> Apheresis, need CBC from Local Lab (in addition to Central Laboratory CBC) | Clarification only, as local CBC needed for safety before proceeding to next day's dose of G-CSF but Central Labs required for data capture purposes. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| Schedule of<br>Events: Post<br>Infusion | Update post busulfan<br>monitoring schedule<br>from every 2 days ±1 to<br>every 3 | Adjusted window allowance for consistency across the 6-week intensive monitoring period to enhance site and subject adherence with the protocol. |
| | days ±1 days, for 6 weeks. Weeks 12, 24, 48 visits-Changed visit window for study visit and associated BM Aspirate and GALT to ±1 week. | Logistical adjustment to better accommodate procedural specialists and study subject availability; enhancing protocol adherence while maintaining reasonable visit and procedural window periods. |
| 6.3.3, 7.1.8,<br>Appendix 4 | Changed text to reflect that Cohort 3 receives two doses of Busulfex over 3 days (Day -4 and Day -2) and how it will be accomplished with real- time, pharmacokineticguided AUC-targeted dosing. | Recommendation of the DSMB from the June 24, 2015 data review meeting to utilize a targeted busulfan dosing strategy (target of 8000 µMol/L*min based on PK of 1 <sup>St</sup> day busulfan infusion) instead of a fixed dose scheme at the 6mg/kg. The AUC target of 8,000 µMol/L*min is recommended by the DSMB as a reduced intensity myeloconditioning regimen derived from experience with busulfan in oncology patients. Updated reference to busulfan visits and dosing in Schedule of Events and throughout document as applicable. |
| 6.3.4 | Changed Post-busulfan infection prophylaxis with trimethoprim-sulfamethoxazole (TMP-SMX) to be administered based on CD4+ T cell count | Due to potential myelosuppressive effects of trimethoprim-sulfamethoxazole (TMP-SMX), changed instructions for administration of TMP-SMX from default administration commencing with busulfan dosing, but rather be based on a subject's risk for Pneumocystis pneumonia (if CD4+ T cell count falls below 200/ml). |
| 7.2.1 | Update post busulfan monitoring schedule from every 2 days ±1 to every 3 days ±1 days, for 6 weeks. | Adjusted window allowance for consistency across the 6-week intensive monitoring period to enhance site and subject adherence with the protocol. |

| <b>Protocol Section</b> | Nature of Change | Rationale |
|---|---|---|
| 7.2.5, Appendix<br>V | Weeks 12, 24, 48 visits-<br>Changed visit windows<br>for study visit and<br>associated<br>BM Aspirate and GALT<br>to<br>±1 week. | Logistical adjustment to better accommodate procedural specialists and study subject availability; enhancing protocol adherence while maintaining reasonable visit and procedural window periods. Updated reference to window periods in Schedule of Events and throughout document as applicable. |
| Administrative/0 | Clerical Updates | |
| Contacts | Update | Integrated an earlier update to the study contacts (version 7.1) into this protocol amendment. |
| 6.3.3 | Changed text to clarify that dose is to be based on subject's weight at the pre-busulfan assessment visit. | Change for clarity only. |
| 7.3 | Changed requirement for creatinine clearance to be estimated by the Cockcroft-Gault equation to now be | The central lab already provides the value utilizing the MDRD equation. This formula does not require the subject's weight to be taken at every visit and is sufficient for this study indication. |
| Appendix 5 | Added wording to allow the autologous plasma collection amounts to be adjusted. | Depending on the cell processing laboratory specifications, these amounts may need to be adjusted for each collection. |
| 6.3.3 | Update "Conditioning<br>Assessment" to "Pre-<br>busulfan Assessment" | Changed to correct visit name. |
| 7.1.5, 7.1.8,<br>7.1.9 | Corrected lab listings to<br>match Schedule of<br>Events | Updated to correct for errors in previous protocol version. |

### **CAL-USA-11: Mock Tables: Table of Contents**

# Contents

| Table 1: Protocol Deviation – Summary | 4 |
|---|---|
| Table 2.1 Protocol Deviation – Major Deviations Summary | 5 |
| Table 2.2 Protocol Deviation – Minor Deviations Summary | |
| Table 3: Demographics and Baseline Information | |
| Table 4: HIV-1 History | |
| Table 5: Manufacturing CD4+ – Cohorts 1 and 2 and 3 | |
| Table 6: Manufacturing CD34 – Cohorts 1 and 2 and 3 | |
| Table 7: Manufacturing Deviations | |
| Table 8.1 Cell Dose (x10e8) at Day 0 vs. Marking/Expression Data | |
| Table 9.1: Busulfan AUC (uMol/min) vs. Marking/Expression Data | 13 |
| Table 10.1: CD4+ Count (mm³) | |
| Table 10.2: CD4+ Count (mm³) vs. Marking/Expression Data | |
| Table 10.3.1. Log <sub>10</sub> HIV-1-RNA Roche Assay (copies/mL) | |
| Table 10.3.2 HIV-1-RNA Abbot Assay (copies/mL) | |
| Table 10.4.1 HIV-1-RNA Roche Assay (copies/mL) vs. Marking/Expression Data | 17 |
| Table 10.4.2 HIV-1-RNA Abbot Assay (copies/mL) vs. Marking/Expression Data | 17 |
| Table 11.1 ANC (10³/uL) vs. Marking/Expression Data | 17 |
| Table 11.2 Platelets (10³/uL) vs. Marking/Expression Data | |
| Table 12 Lymphocyte Development and Chronic Inflammation vs. Marking/Expression | |
| Table 13.1: Adverse Events (Summary SOC, PT) | |
| Table 13.2: Adverse Events by CTC grade (Severity) | 19 |
| Table 13.2: Adverse Events by CTC grade (Severity) (Continued) | |
| Table 13.3: Treatment Emergent Adverse Events by Relationship to Study Drug (Causality) | |
| Table 13.3: Treatment Emergent Adverse Events by Relationship to Study Drug (Causality) | |
| Table 13.4: Treatment Emergent Adverse Events by Relationship to Study Procedure (Causality) | 23 |
| Table 13.4: Adverse Events by Relationship to Study Procedure (Causality) | 24 |

#### **GENERAL COMMENTS**

- Where a count is 0, the percentage will not be shown (e.g. 0(0.0%) will be displayed as 0)
- Unless otherwise states, parameters will be listed in alphabetical order
- Percentages will be presented to one decimal place
- The minimum and maximum values will be presented to the same number of decimal places as recorded in the electronic Case Report Form (eCRF)
- Mean, median, and SD will be presented to one more decimal place than the raw data
- Percentages will be rounded to one decimal place, with the denominator being the number of subjects in the relevant population with non-missing data, unless otherwise specified
- Change from Baseline:

Change from Baseline will be calculated as:

Change from baseline = new value - baseline value

- Unscheduled visits will be excluded from summary tables
- Names and order of Treatment Groups
  - Cohort 1 (No Busulfan)
  - Cohort 2 (One Dose Busulfan)
  - Cohort 3 (Two Dose Busulfan)
  - All
- Names of visits
  - Screening 1
  - Screening 2
  - CD4+ Apheresis
  - G-CSF 1
  - G-CSF 2
  - G-CSF 3
  - G-CSF 4
  - G-CSF 5 + CD34+ Apheresis (For cohorts 1 and 2, CD34 apheresis visit is on the same day as G-CSF 5 (G-CSF 5 + CD34 apheresis). For cohort 3, there are 2 CD34 aphereses: G-CSF 4 & plerixafor + CD34 apheresis & G-CSF 5 + CD34 apheresis)
  - Pre-Busulfan
  - Busulfan (Day -3)
  - Busulfan (Day -2)
  - Infusion (Day 0)
  - Week 1
  - Week 2
  - Week 4
  - Week 6

Strictly 

- Week 8
- Week 12
- Week 16
- Week 20
- Week 24
- Week 32
- Week 40
- Week 48
- Busulfan Follow-up Regimen
- Early Discontinuation
- Follow-up Extension
- Column widths and text-wrapping may be altered in final output to best present the data
- Footnotes may be added/amended if required

Strictly Confidential Page **3** of **24**  Table 1: Protocol Deviation – Summary

Protocol: CAL-USA-11 Population: All Enrolled

| n(%) | Cohort 1<br>(No Busulfan)<br>(N=X) | Cohort 2<br>(One Dose Busulfan)<br>(N=X) | Cohort 3<br>(Two Dose Busulfan)<br>(N=X) | ALL (N=X) |
|---|---|---|---|---|
| Subjects with at least 1 deviation over all | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Number of deviations | X (\(\lambda \lambda \ | X (^^.^/) | X (XA.A/6) | X (XX.X%) |
| Screening 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Screening 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| CD4+ Apheresis | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| G-CSF Administration | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| CD34+ Apheresis | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Busulfan Administration and PK | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| aseline | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Veek 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Veek 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Veek 4 | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |
| Veek 6 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Week 8 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Veek 12 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week 16 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week 20 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Veek 24 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Veek 32 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week 40 | x (xx.x%) | X (XX.X%) | x (xx.x%) | x (xx.x%) |
| Week 48 | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |

Note: Percentage is based on all enrolled subjects.

Clinical cut-off date: DDMMMYYYY

**Programming Note:** This table will be generated from the non-compliance tracker, as provided by the Clin Ops Team.

Strictly Confidential Page **4** of **24**  Table 2.1 Protocol Deviation – Major Deviations Summary

Protocol: CAL-USA-11

Protocol No: CAL-USA-11

Clinical data cut-off date: DDMMMYYYY

**Programming Note:** This table will be prepared by Callimmune.

Table 2.2 Protocol Deviation – Minor Deviations Summary

Protocol: CAL-USA-11

Clinical data cut-off date: DDMMMYYYY

**Programming Note:** This table will be prepared by Callimmune.

Table 3: Demographics and Baseline Information

Protocol: CAL-USA-11
Population: All Enrolled

| n(%) | Cohort 1<br>(No Busulfan) | Cohort 2<br>(One Dose Busulfan) | Cohort 3<br>(Two Dose Busulfan) | ALL |
|---|---|---|---|---|
| | (N=X) | (N=X) | (N=X) | (N=X) |
| Age (years)* | | | | |
| n | X | X | X | Χ |
| Mean | X.X | X.X | X.X | X.X |
| Median | X.X | X.X | X.X | X.X |
| SD | X.X | X.X | X.X | X.X |
| Min | X | X | X | Χ |
| Max | X | X | X | Х |
| Gender (n%) | | | | |
| Female | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Male | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) |
| Race n(%) | | | | |
| Asian | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Black | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| White | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Ethnicity n(%) | | | | |
| Hispanic/Latino | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Non-Hispanic/Latino | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

<sup>\*</sup>Age calculated at date of informed consent: = Integer(Date at informed consent – date of birth +1)/365.25)

SD: Standard Deviation

Clinical data cut-off date: DDMMMYYYY

Table 4: HIV-1 History Protocol: CAL-USA-11 Population: All Enrolled

| | Cohort 1<br>(No Busulfan) | Cohort 2<br>(One Dose Busulfan) | Cohort 3<br>(Two Dose Busulfan) | ALL<br>(N=X) |
|---|---|---|---|---|
| | (N=X) | (N=X) | (N=X) | |
| owest CD4+ T Lymphocyte Count (c | rells/μl) | | | |
| n | X | X | X | Χ |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.X | XXX.X | XXX.X | XXX.X |
| Min | XXX | XXX | XXX | XXX |
| Max | XXX | XXX | XXX | XXX |
| ighest Plasma HIV-1 Viral Load (cop | pies/mL) | | | |
| n | X | X | X | Χ |
| Mean | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X |
| Median | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.> |
| SD | XXX,XXX.X | XXX,XXX.X | XXX,XXX.X | XXX,XXX.> |
| Min | XXX,XXX | XXX,XXX | XXX,XXX | XXX,XXX |
| Max | XXX,XXX | XXX,XXX | XXX,XXX | XXX,XXX |

SD: Standard Deviation

Clinical data cut-off date: DDMMMYYYY

Table 5: Manufacturing CD4+ – Cohorts 1 and 2 and 3

Protocol: CAL-USA-11 Population: Safety

**Programming Note:** Create this table for all cohorts.

Cohort: Cohort 1 (No Busulfan)

| Subject Number | XX-XXXXX | XX-XXXXX | XX-XXXXX | XX-XXXXX |
|---|---|---|---|---|
| CD4+ Apheresis | | | | |
| Apheresis Volume (L) | x.xx | X.XX | X.XX | X.XX |
| Total number of cells collected | xxx.x | XXX.X | XXX.X | XXX.X |
| (x 10^8 cells) | | | | |
| Age of Subject | XX | XX | XX | XX |
| (at Apheresis visit) (yrs) | | | | |
| % of CD4+ in the collected cells | XX.X | XX.X | XX.X | XX.X |
| (% CD4+) | | | | |
| Total number of CD4+ cells collected | XX.X | XX.X | XX.X | XX.X |
| (x 10^8 CD4+) | | | | |
| D4+ Final Cell Product (T <sup>tn</sup> ) | | | | |
| Total viable CD4+ cells | XX.X | XX.X | XX.X | XX.X |
| (At the end of the manufacturing process) | | | | |
| (x 10^8 cells) | | | | |
| Purity (% CD4+) | XX.X | XX.X | XX.X | XX.X |
| Viability (%) | XX.X | XX.X | XX.X | XX.X |
| Transduction Efficiency | XX.X | XX.X | XX.X | XX.X |
| (determined by FACS) (%) | | | | |
| Transduction Efficiency | X.XX | X.XX | X.XX | X.XX |
| (determined by WPRE qPCR) (vector/cell) | | | | |
| Estimated T <sup>tn</sup> Dose | XX.X | XX.X | XX.X | XX.X |
| (based on Body Weight at Apheresis visit) (x 10^6 cells/kg) | | | | |
| nfusion (Baseline) | | | | |
| Body Weight | XXX.X | xxx.x | XXX.X | xxx.x |
| (at Baseline visit) (kg) | **** | ^^.^ | ^^.^ | ^^.^ |
| Actual Ttn Dose | XX.X | XX.X | XX.X | XX.X |
| (based on Body Weight on the Day of Infusion) | AA.A | AA.A | ۸۸.۸ | ^^.^ |
| (x 10 <sup>6</sup> cells/kg) | | | | |

Clinical data cut-off date: DDMMMYYYY

Table 6: Manufacturing CD34 – Cohorts 1 and 2 and 3

Protocol: CAL-USA-11 Population: Safety

**Programming Note:** Create this table for all cohorts.

Cohort: Cohort 1 (No Busulfan)

| Subject Number | XX-XXXXX | XX-XXXXX | XX-XXXXX | XX-XXXXX |
|---|---|---|---|---|
| CD34+ Apheresis | | | | |
| Apheresis Volume (L) | x.xx | X.XX | X.XX | X.XX |
| Total number of cells collected | XXX.X | XXX.X | XXX.X | XXX.X |
| (x 10^8 cells) | | | | |
| Age of Subject | XX | XX | XX | XX |
| (at Apheresis visit) (yrs) | | | | |
| % of CD34+ in the collected cells | XX.X | XX.X | XX.X | XX.X |
| (% CD34+) | | | | |
| Total number of CD34+ cells collected | XX.X | XX.X | XX.X | XX.X |
| (x 10^8 CD4+) | | | | |
| CD34+ Final Cell Product (HSPC <sup>tn</sup> ) | | | | |
| Total viable CD34+ cells | XX.X | XX.X | XX.X | XX.X |
| (At the end of the manufacturing process) | | | | |
| (x 10^8 cells) | | | | |
| <b>Purity</b> (% CD34+) | XX.X | XX.X | XX.X | XX.X |
| Viability (%) | XX.X | XX.X | XX.X | XX.X |
| Transduction Efficiency | XX.X | XX.X | XX.X | XX.X |
| (determined by FACS) (%) | | | | |
| Transduction Efficiency | X.XX | X.XX | X.XX | X.XX |
| (determined by WPRE qPCR) (vector/cell - day 7 | | | | |
| Estimated HSPC <sup>tn</sup> Dose | XX.X | XX.X | XX.X | XX.X |
| (based on Body Weight at Apheresis visit) (x 10 <sup>6</sup> cells/kg) | | | | |
| nfusion (Possiins) | | | | |
| nfusion (Baseline)<br>Body Weight | VVV V | WW V | WW V | WWW W |
| (at Baseline visit) (kg) | XXX.X | XXX.X | XXX.X | XXX.X |
| Actual HSPC <sup>tn</sup> Dose | XX.X | XX.X | XX.X | XX.X |
| (based on Body Weight on the Day of Infusion) | *** | лл.л | хх.х | **** |
| (x 10^6 cells/kg) | | | | |

Clinical data cut-off date: DDMMMYYYY

Table 7: Manufacturing Deviations

Protocol: CAL-USA-11 Population: Safety

Clinical data cut-off date: DDMMMYYYY

**Programming Note:** This table will be prepared by Callimmune.


15 December 2017

Table 8.1 Cell Dose (x10e<sup>8</sup>) at Day 0 vs. Marking/Expression Data

Protocol: CAL-USA-11 Population: Safety

Parameters: Peripheral Blood

Marking/Expression: Cal-1 Marking (WPRE qPCR) (%)

Cohort 1 (No Busulfan) (N=X)

| | | (, | | |
|---|---|---|---|---|
| | Cell Dose a | t Day 0 (x10e <sup>8</sup> ) | Cal-1 Marking (WPRE qPCR) (% | |
| Subject Number | T <sup>tn</sup> (CD4+) Dose | HSPC <sup>tn</sup> (CD34+) Dose | Peak | Week 48 |
| xx-xxxx | XX.XX | XX.XX | XX.XX | XX.XX |
| xx-xxxx | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX |
| xx-xxxxx | XX.XX | XX.XX | XX.XX | XX.XX |
| 1 | X | Χ | Χ | Х |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.X | XXX.X | XXX.X | XXX.X |
| Min | XXX | XXX | XXX | XXX |
| Max | XXX | XXX | XXX | XXX |
| Cell Dose (x10e <sup>8</sup> ) vs. Peak Cal-1 Marking (WPRE qPCR) (%) | | | | |
| Pearson product-moment correlation | x.xxx | x.xxx | | |
| Spearman correlation coefficient | X.XXX | X.XXX | | |
| Cell Dose (x10e <sup>8</sup> ) vs. Week 48 Cal-1 Marking (WPRE qPCR) | (%) | | | |
| Pearson product-moment correlation | x.xxx | x.xxx | | |
| Spearman correlation coefficient | x.xxx | x.xxx | | |

SD: Standard Deviation; "Not Detectable" Cal-Marking WPRE qPCR) (%) is set to 0.

Subject XX-XXXXX: Peak Cal-1 Marking (WPRE qPCR) (%) collected at Week X. Latest time point used as Week 48: Week X.

Clinical cut-off date: DDMMMYYYY

Program: filepath name, Output: filepath name Created: DDMMMYYYY HH:MM

**Programming Note:** Repeat this table for all cohorts and overall.

This table will also be repeated (below) for all parameters (Peripheral Blood, Peripheral Blood Subsets: monocytes, granulocytes, CD8+ lymphocytes, CD4+ lymphocytes, Bone Marrow and GALT (both locations) and all markings/expression (Cal-1 Marking (WPRE qPCR) (copies/cell), Cal-1 C46 Expression (C46 RTqPCR) (relative expression), Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)).
Table 9.1: Busulfan AUC (uMol/min) vs. Marking/Expression Data

Protocol: CAL-USA-11 Population: Safety

Parameters: Peripheral Blood

Marking/Expression: Cal-1 Marking (WPRE qPCR) (%)

| | Cohort 2<br>(One Dose Busulfan)<br>(N=X) | | | | |
|---|---|---|---|---|---|
| | Busulfan AUC<br>(uMol/min) | Busulfan AUC (uMol/min) | Total Busulfan | Cal-1 Marking (WPRE qPCR) (%) | |
| Subject Number | at Day -4 | at Day -2 | AUC (uMol/min) —<br>(Day -4 + Day -2) | Peak | Week 48 |
| xx-xxxxx | N/A | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | 14// | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | | XX.XX | XX.XX | XX.XX | XX.XX |
| xx-xxxx | | XX.XX | XX.XX | XX.XX | XX.XX |
| n | | Χ | X | Х | Х |
| Mean | | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | | XXX.X | XXX.X | XXX.X | XXX.X |
| Min | | XXX | XXX | XXX | XXX |
| Max | | XXX | XXX | XXX | XXX |
| Busulfan AUC (uMol/min)at Day -2 vs. Peak Cal-1 Marking (WPRE qPCR) (%) | | | | | |
| Pearson product-moment correlation | | x.xxx | X.XXX | | |
| Spearman correlation coefficient | | X.XXX | x.xxx | | |
| Busulfan AUC (uMol/min)at Day -2 vs. Week 48 Cal-1 Marking (WPRE qPCR) (%) | | | | | |
| Pearson product-moment correlation | | x.xxx | X.XXX | | |
| Spearman correlation coefficient | | x.xxx | X.XXX | | |

SD: Standard Deviation; "Not Detectable" Cal-Marking WPRE qPCR) (%) is set to 0.

Subject XX-XXXXX: Peak Cal-1 Marking (WPRE qPCR) (%) collected at Week X. Latest time point used as Week 48: Week X.

Clinical cut-off date: DDMMMYYYY
Program: filepath name, Output: filep

#### **Programming Note:**

This table will be repeated (below) for all parameters (Peripheral Blood, Peripheral Blood Subsets: monocytes, granulocytes, CD8+ lymphocytes, CD4+ lymphocytes, Bone Marrow and GALT (both locations) and all markings/expression (Cal-1 Marking (WPRE qPCR) (copies/cell), Cal-1 C46 Expression (C46 RTqPCR) (relative expression), Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)).


Table 10.1: CD4+ Count (mm<sup>3</sup>)

Protocol: CAL-USA-11 Population: Safety

> Cohort 1 (No Busulfan) (N=X)

15 December 2017

Subject Number

| | Baseline | CD4+ Count | t (mm³) | Maxir | num CD4+ Coun<br>transduc | t (mm³) post the<br>ed cell infusion | start of the | Week 48 CD4+ Count (mm³) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Pre-<br>Apheresis | Pre-<br>Infusion | Actual<br>Value | Change from<br>Screening | Change from<br>Pre-Apheresis | Change from<br>Pre-Infusion | Actual<br>Value | Change from<br>Screening | Change from<br>Pre-Apheresis | Change from<br>Pre-Infusion |
| xx-xxxx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| n | Х | Х | X | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Max | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| H <sub>0</sub> : Change = 0<br>95% CI for the Mean<br>P-value (Student t)- | | | | | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX |
| 95% CI for the Median<br>P-value (Signed Rank)- | | | | | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX | (XX.XX, XX.XX)<br>X.XXXX |

SD: Standard Deviation

CD4+ Count (mm3) at Screening = Average of Screening 1 and Screening 2 values

CI: Confidence Interval

Subject XX-XXXXX: Maximum value post the start of the transduced cell infusion collected at Week X. Latest time point used as Week 48: Week X.

Clinical cut-off date: DDMMMYYYY

Classification Strictly 


Table 10.2: CD4+ Count (mm<sup>3</sup>) vs. Marking/Expression Data

Protocol: CAL-USA-11 Population: Safety

Parameters: Peripheral Blood

Marking/Expression: Cal-1 Marking (WPRE qPCR) (%)

Cohort 1

15 December 2017

| | | | | | | | Conort 1 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cultinat Number | | | | | | (1) | lo Busulfan) | | | | | | |
| Subject Number | | | | | CD | 1+ Count (m | (N=X) | | | | | | |
| | | | | | CD2 | 4+ Count (m | im <sup>s</sup> ) | | | | | Cal 1 I | Mankina |
| | Baseline | | | Maxii | mum value | post the sta | irt of the | | 14/6 | ek 48 | | | Marking |
| | | Baseiine | | | transduced cell infusion - | | | | VVE | | (WPRE qPCR) (%) | | |
| | | | | | Change | Change | Change | | Change | Change | Change | | |
| | | Pre- | Pre- | Actual | from | from Pre- | from Pre- | Actual | from | from Pre- | from Pre- | | |
| | Screening | Apheresis | Infusion | Value | Screening | Apheresis | Infusion | Value | Screening | Apheresis | Infusion | Peak | Week 48 |
| xx-xxxx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX-XXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| N. N | 70.070 | 700000 | 70000 | 701.701 | 701.701 | 700701 | 70.070 | 7011701 | 70.070 | 701701 | 701.701 | 7000 | 7011701 |
| n | Χ | Χ | Χ | Х | Χ | Χ | Χ | X | Χ | Х | Χ | Χ | Χ |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Max | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| CD4+ Count (mm³) vs. Peak Cal-1<br>Marking (WPRE qPCR) (%)<br>Pearson product-moment correlation | x.xxx | x.xxx | x.xxx | | x.xxx | x.xxx | x.xxx | | x.xxx | x.xxx | x.xxx | | |
| Spearman correlation coefficient | X.XXX | X.XXX | X.XXX | | X.XXX | X.XXX | x.xxx | | X.XXX | X.XXX | X.XXX | | |
| CD4+ Count (mm³) vs. Week 28 Cal-1<br>Marking (WPRE qPCR) (%)<br>Pearson product-moment correlation<br>Spearman correlation coefficient | x.xxx<br>x.xxx | x.xxx<br>x.xxx | x.xxx<br>x.xxx | | x.xxx<br>x.xxx | X.XXX<br>X.XXX | x.xxx<br>x.xxx | | x.xxx<br>x.xxx | X.XXX<br>X.XXX | x.xxx<br>x.xxx | | |

Strictly Confidential Page **15** of **24**  SD: Standard Deviation; "Not Detectable" Cal-Marking WPRE qPCR) (%) is set to 0. CD4+ Count (mm<sup>3</sup>) at Screening = Average of Screening 1 and Screening 2 values

Subject XX-XXXXX: Maximum CD4+ Count (mm³) value post the start of the transduced cell infusion collected at Week X. Latest time point used as Week 48: Week X. Peak Cal-1 Marking (WPRE qPCR) (%) collected at Week X. Latest time point used as Week 48: Week X.

Clinical cut-off date: DDMMMYYYY

Program: filepath name, Output: filepath name Created: DDMMMYYYY HH:MM

**Programming Note:** Repeat this table for all applicable cohorts and overall.

This table will also be repeated (below) for all parameters (Peripheral Blood, Peripheral Blood Subsets: monocytes, granulocytes, CD8+ lymphocytes, CD4+ lymphocytes, Bone Marrow and GALT (both locations) and all markings/expression (Cal-1 Marking (WPRE qPCR) (copies/cell), Cal-1 C46 Expression (C46 RTqPCR) (relative expression), Cal-1 sh5 Expression (sh5 RTqPCR) (relative expression)).

Strictly 

#### Table 10.3.1. Log<sub>10</sub> HIV-1-RNA Roche Assay (copies/mL)

Repeat Table 10.1, but include minimum Log<sub>10</sub> HIV-1-RNA Roche Assay value post the start of the transduced cell infusion, not maximum Log<sub>10</sub> HIV-1-RNA Roche Assay value.

#### Table 10.3.2 HIV-1-RNA Abbot Assay (copies/mL)

Repeat Table 10.1, but include minimum Log<sub>10</sub> HIV-1-RNA Roche Assay value post the start of the transduced cell infusion, not maximum Log<sub>10</sub> HIV-1-RNA Abbot Assay value.

#### Table 10.4.1 HIV-1-RNA Roche Assay (copies/mL) vs. Marking/Expression Data

Repeat Table 10.2, but include minimum Log<sub>10</sub> HIV-1-RNA Roche Assay value post the start of the transduced cell infusion, not maximum Log<sub>10</sub> HIV-1-RNA Roche Assay value.

#### Table 10.4.2 HIV-1-RNA Abbot Assay (copies/mL) vs. Marking/Expression Data

Repeat Table 10.2, but include minimum Log<sub>10</sub> HIV-1-RNA Roche Assay value post the start of the transduced cell infusion, not maximum Log<sub>10</sub> HIV-1-RNA Abbot Assay value.

#### Table 11.1 ANC (10<sup>3</sup>/uL) vs. Marking/Expression Data

Repeat Table 10.2, but include minimum ANC value post the start of the transduced cell infusion, not maximum ANC value.

#### Table 11.2 Platelets (10<sup>3</sup>/uL) vs. Marking/Expression Data

Repeat Table 10.2, but include minimum Platelet value post the start of the transduced cell infusion, not maximum Platelet value.

#### Table 12 Lymphocyte Development and Chronic Inflammation vs. Marking/Expression

Repeat Table 10.2 for Lymphocyte Development and Chronic Inflammation parameters

Strictly 

Table 13.1: Adverse Events (Summary SOC, PT)

Protocol: CAL-USA-11 Population: Safety

| | Cohort 1<br>(No Busulfan)<br>(N=X) | | Cohort 2<br>(One Dose Busulfan)<br>(N=X) | | Cohoi<br>(Two Dose I<br>(N=) | Busulfan) | ALL<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Subjects | AEs | Subjects | AEs | Subjects | AEs | Subjects | AEs |
| All Body Systems | X (XX.X%) | Χ | X (XX.X%) | X | 0 | Х | X (XX.X%) | Χ |
| SOC1 | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | Х |
| PT1 | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | Х |
| PT2 | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | X | X (XX.X%) | Χ |
| PTx | <br>X (XX.X%) | <br>X | <br>X (XX.X%) | <br>X | <br>X (XX.X%) | <br>X | <br>X (XX.X%) | <br>X |
| SOC2 | X (XX.X%) | Χ | 0 | Χ | X (XX.X%) | Χ | X (XX.X%) | Χ |
| PT1 | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | X |
| PT2 | X (XX.X%) | Χ | X (XX.X%) | Χ | X (XX.X%) | X | X (XX.X%) | Χ |
| PTx | 0 | Χ | X (XX.X%) | Χ | X (XX.X%) | X | X (XX.X%) | Χ |

AE: Adverse Events

Clinical cut-off date: DDMMMYYYY

Table 13.2: Adverse Events by CTC grade (Severity)

Protocol: CAL-USA-11 Population: Safety

| | | Coho<br>(No Bu:<br>(N= | sulfan) | Cohort 2<br>(One Dose Busulfan)<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Potentially | | | | | |
| | Mild | Moderate | Severe | Life- | Mild | Moderate | Severe | Life- |
| System Organ Class (SOC) Preferred Term (PT) | (Grade 1) | (Grade 2) | (Grade 3) | Threatening<br>(Grade 4) | (Grade 1) | (Grade 2) | (Grade 3) | Threatening<br>(Grade 4) |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum severity within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

Table 13.2: Adverse Events by CTC grade (Severity) (Continued)

Protocol: CAL-USA-11 Population: Safety

| | | Coho<br>(Two Dose | | | ALL | | | |
|---|---|---|---|---|---|---|---|---|
| | | ` (N= | =X) | | | (N=X) | | |
| | | | | Potentially | | | Potentially | |
| | Mild | Moderate | Severe | Life- | Mild | Moderate | Severe | Life- |
| System Organ Class (SOC) Preferred Term (PT) | (Grade 1) | (Grade 2) | (Grade 3) | Threatening<br>(Grade 4) | (Grade 1) | (Grade 2) | (Grade 3) | Threatening (Grade 4) |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| •••• | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum severity within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

Table 13.3: Treatment Emergent Adverse Events by Relationship to Study Drug (Causality)

Protocol: CAL-USA-11 Population: Safety

| | | | | Cohort 2 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (No Busulfan) | ) | | (One Dose Busulfan) | | | | |
| | | | (N=X) | | | | (N=X) | | | |
| System Organ Class (SOC) | Not | Doubtful | Possible | Probable | Very Likely | Not | Doubtful | Possible | Probable | Very Likely |
| Preferred Term (PT) | Related | Doubtiui | POSSIBLE | Probable | very Likely | Related | Doubtiui | FOSSIBLE | Probable | very Likely |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum relatedness within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

Table 13.3: Treatment Emergent Adverse Events by Relationship to Study Drug (Causality)

Protocol: CAL-USA-11 Population: Safety

| | | | Cohort 3 | _ | | | | ALL | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (Tw | o Dose Busul | fan) | | | | | | |
| | | | (N=X) | | | | | (N=X) | | |
| System Organ Class (SOC) | Not | Doubtful | Dossible | Droboblo | VomeLikole | Not | Doubtful | Dossible | Droboblo | Many Likaly |
| Preferred Term (PT) | Related | Doubtful | Possible | Probable | Very Likely | Related | Doubtful | Possible | Probable | Very Likely |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| **** | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum relatedness within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

Table 13.4: Treatment Emergent Adverse Events by Relationship to Study Procedure (Causality)

Protocol: CAL-USA-11 Population: Safety

Study Procedure: Busulfan

| | Cohort 1<br>(No Busulfan)<br>(N=X) | | | | | | Cohort 2<br>(One Dose Busulfan)<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class (SOC)<br>Preferred Term (PT) | Not<br>Related | Doubtful | Possible | Probable | Very Likely | Not<br>Related | Doubtful | Possible | Probable | Very Likely |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum relatedness within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat for all study procedures: GCSF, : Bone Marrow Aspiration, etc.

Table 13.4: Adverse Events by Relationship to Study Procedure (Causality)

Protocol: CAL-USA-11 Population: Safety

Study Procedure: Busulfan

| | | | Cohort 3 | | | | | ALL | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (Tw | o Dose Busul | fan) | | | | | | |
| | | | (N=X) | | (N=X) | | | | | |
| System Organ Class (SOC) | Not | Doubtful | Dossible | Drobable | Vom Likoly | Not | Doubtful | Dossible | Droboblo | Vom Likoly |
| Preferred Term (PT) | Related | Doubtful | Possible | Probable | Very Likely | Related | Doubtful | Possible | Probable | Very Likely |
| All Body Systems | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SOC2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PT2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| PTx | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Subjects are counted once at maximum relatedness within each sub grouping

Note: Percentages are based on the number of subjects in each group

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat for all study procedures: GCSF, : Bone

Marrow Aspiration, etc.

## **CAL-USA-11: Mock Listings: Table of Contents**

# Contents

| isting 1.1: Subject Disposition | 5 |
|---|---|
| isting 1.2: Subject Disposition (continued) | <del>(</del> |
| isting 2: Subject Withdrawal | 7 |
| isting 3: Subject Discontinuation | 8 |
| isting 4.1: Demographics | |
| isting 4.2: Pre-Busulfan Body Weight | 10 |
| isting 5: HIV-1 History | 11 |
| isting 6: Medical History | 12 |
| isting 7: Eligibility | 13 |
| isting 8.1: Pregnancy Test | |
| isting 8.2: Positive Pregnancy Test | 15 |
| isting 9: Chest X-Rays | 16 |
| isting 10: ART Therapy History (regimen overview) | |
| isting 11: Transduced CD4+ Cell Product Dose (Transduction efficiency, viability, cell numbers for T <sup>tn</sup> ) | 18 |
| isting 12: Transduced CD34+ Cell Product Dose (Transduction efficiency, viability, cell numbers for HSPC <sup>tn</sup> ) | 19 |
| isting 13.1: G-CSF Therapy | 20 |
| isting 13.2: Plerixafor Therapy | 21 |
| isting 14.1: Apheresis - CD4+ | |
| isting 14.2: Apheresis - CD34+ | 23 |
| isting 15.1: Busulfan Dosing | 24 |
| isting 15.1: Busulfan Interruptions | 25 |
| isting 15.3: Busulfan Administration and Pharmacokinetics | |
| isting 16: Cal-1 Marking/Expression - Peripheral Blood | |
| isting 17: Cal-1 Marking/Expression – Bone Marrow | 28 |
| isting 18: Cal-1 Marking/Expression – GALT | |
| isting 19.1: Cal-1 Marking/Expression – Subsets Monocytes | |
| isting 19.2: Cal-1 Marking/Expression – Subsets: Granulocytes | |
| isting 19.3: Cal-1 Marking/Expression – Subsets: CD4+ Lymphocytes | |
| isting 19.4: Cal-1 Marking/Expression – Subsets: CD8+ Lymphocytes | |
| isting 20.1: Serious Adverse Events, including event narratives | |
| isting 20.2: Deaths | |
| isting 21.1: Adverse Events (All Grades) | |
| isting 21.2: Adverse Events (Grades 3 and /or 4) | 37 |

| Listing 21.3: Related Adverse Events (Grades 3 and /or 4) | 38 |
|-----------------------------------------------------------|----|
| Listing 22.1: Concomitant Medication | 39 |
| Listing 22.2: Concomitant Procedures and Therapies | 40 |
| Listing 23.1: Laboratory – Hematology | |
| Listing 23.2: Laboratory – Hematology (Abnormal only) | 42 |
| Listing 24.1: Laboratory – Biochemistry | 43 |
| Listing 24.2: Biochemistry (Abnormal only) | |
| Listing 25.1: Lymphocyte phenotype | 45 |
| Listing 25.2: Thymopoieisis | 46 |
| Listing 25.3: Inflammation | 47 |
| Listing 25.4: Maturation | 48 |
| Listing 26: Laboratory – HIV-1 RNA | |
| Listing 27.1: Vital Signs | 50 |
| Listing 27.2: Abnormal Vital Signs | |
| Listing 28.1: Physical Examination | 52 |
| Listing 28.2: Abnormal: Physical Examination | 53 |
| Listing 29.1: Cal-1 Integration Analysis | 54 |
| Listing 29.2: Cal-1 Integration Analysis (Re-test) | |
| Listing 30: Replication Competent Lentivirus (RCL) | 56 |
| Listing 31: HIV-1 Tropism Assay | 57 |
| Listing 32.1: C46 Immunogenicity – Humoral Response | 58 |
| licting 32.2: CA6 Immunogenicity — Cellular Response | 50 |

### **GENERAL COMMENTS**

- Names and order of Treatment Groups
  - Cohort 1 (No Busulfan)
  - Cohort 2 (One Dose Busulfan)
  - Cohort 3 (Two Dose Busulfan)
  - All
- Names of visits
  - Screening 1
  - Screening 2
  - CD4+ Apheresis
  - G-CSF 1
  - G-CSF 2
  - G-CSF 3
  - G-CSF 4
  - G-CSF 5 + CD34+ Apheresis (For cohorts 1 and 2, CD34 apheresis visit is on the same day as G-CSF 5 (G-CSF 5 + CD34 apheresis). For cohort 3, there are 2 CD34 aphereses: G-CSF 4 & plerixafor + CD34 apheresis & G-CSF 5 + CD34 apheresis)
  - Pre-Busulfan
  - Busulfan (Day -3)
  - Busulfan (Day -2)
  - Infusion (Day 0)
  - Week 1
  - Week 2
  - Week 4
  - Week 6
  - Week 8
  - Week 12
  - Week 16
  - Week 20
  - Week 24
  - Week 32
  - Week 40
  - Week 48
  - Busulfan Follow-up Regimen
  - Early Discontinuation


- Follow-up Extension
- Column widths and text-wrapping may be altered in final output to best present the data
- Footnotes may be added/amended if required


Listing 1.1: Subject Disposition

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Informed<br>Consent Date<br>(YYYY-MM-DD) | CD34+<br>Apheresis Date<br>(YYYY-MM-DD) | Infusion Date<br>(YYYY-MM-DD) | Enrolled Population | Safety Population |
|---|---|---|---|---|---|
| xx-xxxxxx | YYYY-MM-DD | YYYY-MM-DD | YYYY-MM-DD | Yes | No |
| xx-xxxxx | YYYY-MM-DD | YYYY-MM-DD | YYYY-MM-DD | Yes | No |
| xx-xxxxxx<br>xx-xxxxxx | YYYY-MM-DD<br>YYYY-MM-DD | YYYY-MM-DD<br>YYYY-MM-DD | YYYY-MM-DD<br>YYYY-MM-DD | Yes<br>Yes | Yes<br>Yes |

Clinical cut-off date: DDMMMYYYY

Listing 1.2: Subject Disposition (continued)

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | CD4+<br>Apheresis Date<br>(YYYY-MM-DD) | Status (Ongoing,<br>Discontinuation,<br>Withdrawal or<br>Completion) <sup>1</sup> | Date of Discontinuation, Withdrawal or Completion (YYYY-MM-DD) | Date Antiretroviral<br>Therapy<br>Commenced | Time from CD4+ Apheresis to Commencement of ART (days) <sup>3</sup> | Last Visit<br>Prior to<br>Discontinuation<br>or Withdrawal | Last<br>Scheduled<br>Visit | Primary Reason for<br>Discontinuation or<br>Withdrawal2 |
|---|---|---|---|---|---|---|---|---|
| XX-XXXXXX | YYYY-MM-DD | Discontinuation | YYYY-MM-DD | YYYY-MM-DD | xx | Week xx | Week xx | Commencement of antiretroviral therapy |
| XX-XXXXXX | YYYY-MM-DD | Discontinuation | YYYY-MM-DD | | xx | Week xx | Week xx | Commencement of antiretroviral therapy |
| XX-XXXXXX<br>XX-XXXXXX | YYYY-MM-DD<br>YYYY-MM-DD | Completed<br>Completed | YYYY-MM-DD<br>YYYY-MM-DD | | xx<br>xx | -<br>- | Week xx<br>Week xx | and ed ornal therapy |

<sup>&</sup>lt;sup>1</sup> Withdrawal: any subject who withdrew consent from the trial; Discontinuation: any subject who discontinued from primary endpoint analysis <sup>2</sup> Last scheduled visit before discontinuation or withdrawal.

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Include all detail with regards to reason for discontinuation in "Primary Reason for Discontinuation or Withdrawal<sup>2</sup>":

- SAE number if applicable
- AE number if applicable
- Manufacturing failure details if applicable

<sup>&</sup>lt;sup>3</sup> Date Antiretroviral Therapy Commenced / Date of Discontinuation, Withdrawal or Completion - CD4+ Apheresis Date + 1

Listing 2: Subject Withdrawal

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject Number | Date of Withdrawal<br>(YYYY-MM-DD) | Phase of<br>Withdrawal <sup>1</sup> | Primary Reason for Withdrawal | Secondary Reason for Withdrawal * |
|---|---|---|---|---|
| (X-XXXXX<br>(X-XXXXXX<br>(X-XXXXXX | YYYY-MM-DD<br>YYYY-MM-DD<br>YYYY-MM-DD | Post-infusion phase | Commencement of antiretroviral therapy | Other: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Clinical cut-off date: DDMMMYYYY

<sup>\*</sup> Withdrawal occurred in Post-Infusion phase.

<sup>1</sup> Withdrawal: any subject who withdrew consent from the trial

Listing 3: Subject Discontinuation

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | Date of Discontinuation | Phase of | Last Visit Prior to | |
|---|---|---|---|---|
| Subject Number | (YYYY-MM-DD) | Discontinuation | Discontinuation | Primary Reason for Discontinuation |
| xx-xxxxx | YYYY-MM-DD | Post-infusion phase | Week xx | Commencement of antiretroviral therapy |
| XX-XXXXX | YYYY-MM-DD | Post-infusion phase | Week xx | Commencement of antiretroviral therapy |
| xx-xxxxx | YYYY-MM-DD | Post-infusion phase | Week xx | Commencement of antiretroviral therapy |

Note: Subject discontinuation refers to any subject who discontinued from the primary endpoint analysis

Clinical cut-off date: DDMMMYYYY

Listing 4.1: Demographics Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Center | Gender | Date of Birth<br>(YYYY-MM-DD) | Age* | Race | Ethnicity | Child Bearing Potential |
|---|---|---|---|---|---|---|---|
| XX-XXXXXX<br>XX-XXXXXX | Quest Clinical Research: Dr Lalezari<br>UCLA CARE Center Clinic: Dr | Male<br>Male | YYYY-MM-DD<br>YYYY-MM-DD | XX<br>XX | White<br>White | Not Hispanic or Not Latino<br>Not Hispanic or Not Latino | |
| xx-xxxxxx | Mitsuyasu<br>Quest Clinical Research: Dr Lalezari | Female | YYYY-MM-DD | xx | White | Not Hispanic or Not Latino | Yes |

<sup>\*</sup> Age calculated at date of informed consent

Clinical cut-off date: DDMMMYYYY

Strictly Confidential Page **9** of **59**  Listing 4.2: Pre-Busulfan Body Weight

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 2

| Subject<br>Number | Date Performed<br>(YYYY-MM-DD) | Time Performed<br>(HH:MM) | Actual Weight (kg) | Adjusted ideal body weight<br>(AIBW) | Was Actual Weight OR<br>adjusted ideal body weight<br>(AIBW) used for the Calculation<br>of the Busulfan dose |
|---|---|---|---|---|---|
| xx-xxxxx | YYYY-MM-DD | HH:MM | XX.X | XX.X | Actual Weight |
| XX-XXXXXX | YYYY-MM-DD | HH:MM | xx.x | xx.x | Actual Weight |
| XX-XXXXX | YYYY-MM-DD | HH:MM | xx.x | xx.x | Actual Weight |
| XX-XXXXXX | YYYY-MM-DD | HH:MM | xx.x | xx.x | Actual Weight |
| XX-XXXXXX | YYYY-MM-DD | HH:MM | XX.X | xx.x | Actual Weight |

Clinical cut-off date: DDMMMYYYY


Listing 5: HIV-1 History Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject Number | Date of HIV-1 infection<br>Diagnosis<br>(YYYY-MM-DD) | Lowest CD4+<br>T Lymphocyte Count<br>(cells/µl) | Date of Lowest CD4+<br>Count<br>(YYYY-MM-DD) | Highest Plasma HIV Viral<br>Load<br>(copies/mL) | Date of Highest HIV Viral<br>Load<br>(YYYY-MM-DD) |
|---|---|---|---|---|---|
| XX-XXXXX | YYYY-MM-DD | XXX | YYYY-MM-DD | XXXXXXX | YYYY-MM-DD |
| XX-XXXXXX | YYYY-MM-DD | xxx | YYYY-MM-DD | xxxxxxx | YYYY-MM-DD |
| XX-XXXXXX | YYYY-MM-DD | XXX | YYYY-MM-DD | XXXXXXX | YYYY-MM-DD |

NK: Not Known

Clinical cut-off date: DDMMMYYYY

Listing 6: Medical History Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject | MH | | Onset Date | Resolution Date | | Any Treatment |
|---|---|---|---|---|---|---|
| Number | No Condition | Body System Code | (YYYY-MM-DD) | (YYYY-MM-DD) | Ongoing? | Planned? |
| xx-xxxxxx | 1 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Dermatologic | YYYY-MM-DD | | Yes | No |
| | 3 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Neurological | YYYY-MM-DD | YYYY-MM-DD | No | No |
| | 4 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Other: fainting | YYYY-MM-DD | YYYY-MM-DD | No | No |
| | 6 xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Allergies/Drug Sensitivity | NK | | Yes | No |
| | Etc. | | | | | |
| xx-xxxxx | X xxxxxxxxxxxxxxxxxxxxxxx | Ears | NK | | Yes | No |

NK: Not Known; MH No: Medical History Number

Clinical cut-off date: DDMMMYYYY


Listing 7: Eligibility
Protocol: CAL-USA-11
Population: All Screened

Cohort: Cohort 1

| | | | Inclusion Criteria | | Exclusion Criteria |
|---|---|---|---|---|---|
| Subject<br>Number | Evaluation Date<br>(YYYY-MM-DD) | Criteria<br>Not Met* | Reason Not Met | Criteria<br>Met* | Reason Met |
| XX-XXXXXX | YYYY-MM-DD | xxxxx | HIV-1 VIRAL RNA LESS THAN 5000 COPIES/ML | | |
| XX-XXXXXX | YYYY-MM-DD | XXXXX | screening cd4 <500 | XXXXX | cd4 history <250 |
| xx-xxxxxx | YYYY-MM-DD | xxxxx | Plasma HIV-1 viral RNA < 5,000 copies/ml reported on August 31, 2013 | | |
| xx-xxxxxx | YYYY-MM-DD | xxxxx | CD4 <500 | | |
| xx-xxxxxx | YYYY-MM-DD | xxxxx | HIV-1 RNA > 100,000 copies/ml at Screen 1 reported on December 29, 2013 | | |
| xx-xxxxxx | YYYY-MM-DD | xxxxx | viral load 190,000 | | |
| xx-xxxxx | YYYY-MM-DD | xxxxx | CD4+ T lymphocyte count < 500 at Screen 2 reported on September 18, 2013" | | |

<sup>\*</sup> Inclusion & Exclusion Criteria: refer to Protocol CAL-USA-11, Section 5

Clinical cut-off date: DDMMMYYYY

Listing 8.1: Pregnancy Test Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Visit | Date of<br>Collection<br>(YYYY-MM-DD) | Time of<br>Collection<br>(HH:MM) | Variable*<br>(Serum ß-HCG or<br>Urine Test) | Result | Unit | Clin Sig.** | Comment |
|---|---|---|---|---|---|---|---|---|
| xx-xxxxxx | Screening 1 | YYYY-MM-DD | HH:MM | xxxxxxxxxxxx | Negative | xxxxx | | xxxxxxxxxx |
| | Screening 2 | YYYY-MM-DD | HH:MM | xxxxxxxxxxxx | Negative | XXXXX | | XXXXXXXXXX |
| | G-CSF-1 | YYYY-MM-DD | HH:MM | XXXXXXXXXXXX | Negative | xxxxx | | xxxxxxxxxx |
| (X-XXXXX | | | | | | | | |
| (X-XXXXXX | | | | | | | | |

<sup>\*</sup> Serum ß-HCG testing from women of reproductive potential, except at commencement of G-CSF, busulfan and infusion (baseline), when urine test is performed \*\* Clinical Significance: CS=Clinically Significant, NCS=Not Clinically Significant

Clinical cut-off date: DDMMMYYYY

15 December 2017


Listing 8.2: Positive Pregnancy Test

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Visit | Date of<br>Collection<br>(YYYY-MM-DD) | Time of<br>Collection<br>(HH:MM) | Variable*<br>(Serum ß-HCG or<br>Urine Test) | Result | Unit | Clin Sig.** | Comment |
|---|---|---|---|---|---|---|---|---|
| XX-XXXXXX | Screening 1 | YYYY-MM-DD | HH:MM | xxxxxxxxxxxx | Positive | xxxxx | NCS | xxxxxxxxxx |
| | Screening 2 | YYYY-MM-DD | HH:MM | XXXXXXXXXXXXX | Positive | XXXXX | NCS | XXXXXXXXXX |
| | G-CSF-1 | YYYY-MM-DD | HH:MM | XXXXXXXXXXXX | Positive | xxxxx | NCS | xxxxxxxxx |

XX-XXXXX XX-XXXXXX

Clinical cut-off date: DDMMMYYYY

<sup>\*</sup> Serum ß-HCG testing from women of reproductive potential, except at commencement of G-CSF, busulfan and infusion (baseline), when urine test is performed \*\* Clinical Significance: CS=Clinically Significant, NCS=Not Clinically Significant

Listing 9: Chest X-Rays Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| ubject<br>Iumber | Visit | Date Performed<br>(YYYY-MM-DD) | Result (If CS, specify)* |
|---|---|---|---|
| x-xxxxx | Screening 1 | YYYY-MM-DD | Normal |
| | Screening 2 | YYYY-MM-DD | Abnormal – NCS |
| -xxxxx | Screening 1 | YYYY-MM-DD | Norma; |
| | Screening 2 | YYYY-MM-DD | Normal |

<sup>\*</sup>Clinical Significance: CS=Clinically Significant, NCS=Not Clinically Significant

Clinical cut-off date: DDMMMYYYY

Listing 10: ART Therapy History (regimen overview)

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | Regimen | | Start Date | Stop Date | | Reason for<br>Discontinuation | Lowest Plasma HIV Viral Load<br>Achieved During Regimen |
|---|---|---|---|---|---|---|---|
| Subject Number | Number | Drug | (YYYY-MM-DD) | (YYYY-MM-DD) | Ongoing | of therapy | (copies/mL) |
| xx-xxxxx | 1 | 3ТС | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <500 |
| | | D4T | YYYY-MM-DD | YYYY-MM-DD | No | , | |
| | | INVIRASE | YYYY-MM-DD | YYYY-MM-DD | No | | |
| | 2 | CRIXIVAN | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <500 |
| | | COMBIVIR | YYYY-MM-DD | YYYY-MM-DD | No | , | |
| | 3 | COMBIVIR | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <50 |
| | | SUSTIVA | YYYY-MM-DD | YYYY-MM-DD | No | 3 | |
| XX-XXXXX | 1 | Complera | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <20 |
| (X-XXXXX | 1 | ATRIPLA | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <20 |
| | 2 | COMPLERA | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <20 |
| X-XXXXX | 1 | truvada | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <20 |
| | | isentress | YYYY-MM-DD | YYYY-MM-DD | No | S | |
| XX-XXXXX | 1 | Miraviroc | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <50 |
| | 2 | Atripla | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <75 |
| | 3 | complera | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <75 |
| XX-XXXXX | 1 | stribild | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <20 |
| | 2 | stribild | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | 44 |
| XX-XXXXX | 1 | ISENTRESS | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <20 |
| | | TRUVADA | YYYY-MM-DD | YYYY-MM-DD | No | _ | |
| XX-XXXXX | 1 | truvada | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | <40 |
| | | miraviroc | YYYY-MM-DD | YYYY-MM-DD | No | • | |
| | 2 | darunavir | YYYY-MM-DD | YYYY-MM-DD | No | Toxicity | unk |
| | | ritonavir | YYYY-MM-DD | YYYY-MM-DD | No | • | |
| | 3 | truvada | YYYY-MM-DD | YYYY-MM-DD | No | Treatment fatigue | <40 |
| | | raltegravir | YYYY-MM-DD | YYYY-MM-DD | No | S | |

NK: Not Known

Clinical cut-off date: DDMMMYYYY

Listing 11: Transduced CD4+ Cell Product Dose (Transduction efficiency, viability, cell numbers for T<sup>tn</sup>)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | - | Total Number of Cells Infused <sup>1</sup> | | | | | |
|---|---|---|---|---|---|---|---|
| | Date of TCP<br>Infusion<br>(YYYY-MM-DD) | Absolute<br>(x10 <sup>8</sup> cells) | Expressed as<br>cells/kg body weight<br>(x10 <sup>6</sup> cells/kg) | Viability<br>(%)² | Purity of cells infused | Transduction Efficiency of<br>Cells Infused (%) | Cal-1 Vector Copy Number<br>(VCN) per T <sup>tn</sup> cell (VCN/cell) |
| XX-XXXXXX | YYYY-MM-DD | xx | XX.X | xx | xx.x | XX.X | XX.X |
| XX-XXXXXX | YYYY-MM-DD | XX | xx.x | XX | XX.X | xx.x | xx.x |
| XX-XXXXX | YYYY-MM-DD | XX.X | xx.x | XX.X | XX.X | xx.x | xx.x |
| XX-XXXXXX | YYYY-MM-DD | XX.X | XX.X | XX | XX.X | XX.X | XX.X |

<sup>&</sup>lt;sup>1</sup> Viable, transduced cells (viability based on pre-thaw viability)

TCP: Transduced Cell Product

Clinical cut-off date: DDMMMYYYY

Program: filepath name, Output: filepath name Created: DDMMMYYYY HH:MM


<sup>&</sup>lt;sup>2</sup> Pre-thaw viability of T<sup>tn</sup> cells (%)

T<sup>tn</sup>: Cal-1 transduced CD4+ T lymphocytes

Listing 12: Transduced CD34+ Cell Product Dose (Transduction efficiency, viability, cell numbers for HSPC<sup>tn</sup>)

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | _ | Total Number of Cells Infused <sup>1</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Date of TCP<br>Infusion<br>(YYYY-MM-DD) | Absolute<br>(x10 <sup>8</sup> cells) | Expressed as<br>cells/kg body<br>weight<br>(x10 <sup>6</sup> cells/kg) | Viability<br>(%)² | Purity of cells<br>infused | Transduction Efficiency of Cells Infused (%) | Cal-1 Vector Copy<br>Number (VCN) per Ttn<br>cell (VCN/cell) | Was the CD34+<br>back-up apheresis<br>product infused |
| | \/\/\/\ NANA DD | | | | | | | |
| XX-XXXXXX | YYYY-MM-DD | XX | XX.X | XX | XX.X | XX.X | XX.X | - |
| XX-XXXXX | YYYY-MM-DD | XX | XX.X | XX | XX.X | XX.X | XX.X | - |
| XX-XXXXX | YYYY-MM-DD | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | - |
| XX-XXXXX | YYYY-MM-DD | XX.X | XX.X | XX | XX.X | XX.X | xx.x | - |
| | | | | | | | | - |

<sup>&</sup>lt;sup>1</sup> Viable, transduced cells (viability based on pre-thaw viability) <sup>2</sup> Pre-thaw viability of HSPC<sup>tn</sup> cells (%)

TCP: Transduced Cell Product

HSPC<sup>tn</sup>: Cal-1 transduced CD34+ Hematopoietic stem/progenitor cells

Clinical cut-off date: DDMMMYYYY


Listing 13.1: G-CSF Therapy Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | | Dose | Total Daily<br>Dose | | | Time Second Dose | Was the White blood cell count on Day 4 |
|---|---|---|---|---|---|---|---|---|
| Subject | | Was G-CSF | Administered | Administered | Full Dose | Date/ Time Administered | Administered | of G-CSF < |
| Number | Visit | Administered? | (μg/kg) | (μg) | Administered? | (YYYY-MM-DD) / HH:MM | HH:MM | 75,000x10e9/mL? |
| XX-XXXXX | G-CSF 1 | Yes | 10μg/kg QD | XXX | - | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 2 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 3 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 4 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | CD34+ Apheresis | | | | | | | XX |
| XX-XXXXXX | G-CSF 1 | Yes | 10μg/kg QD | xxx | _ | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 2 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 3 | Yes | 10μg/kg QD | _ | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 4 | Yes | 10μg/kg QD | _ | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | CD34+ Apheresis | . 65 | 10 MO/ 118 Q1 | | . 00 | 227 | | XX |
| xx-xxxxxx | G-CSF 1 | Yes | 10μg/kg QD | xxx | _ | YYYY-MM-DD/ HH:MM | HH:MM | |
| ********* | G-CSF 2 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 3 | Yes | 10μg/kg QD | _ | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 4 | Yes | 10μg/kg QD<br>10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | | 163 | τυμg/ kg QD | - | 165 | אוואוואו לסמי-ואוואו | TITI.IVIIVI | VV |
| | CD34+ Apheresis | | | | | | | XX |
| XX-XXXXXX | G-CSF 1 | Yes | 10μg/kg QD | xxxxx | - | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 2 | Yes | 10μg/kg QD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 3 | Yes | 5μg/kg BD | - | No | YYYY-MM-DD/ HH:MM | HH:MM | |
| | G-CSF 4 | Yes | 5μg/kg BD | - | Yes | YYYY-MM-DD/ HH:MM | HH:MM | |
| | CD34+ Apheresis | | . 5. 0 | | | · | | XX |

Clinical cut-off date: DDMMMYYYY

Listing 13.2: Plerixafor Therapy

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 3

| le i e et | | Total Daily Dose | Data / Time a Advantage to your |
|---|---|---|---|
| ubject | | Administered | Date/ Time Administered |
| lumber | Visit | (μg) | (YYYY-MM-DD) / HH:MM |
| x-xxxxx | G-CSF 4 & plerixafor | xxx | YYYY-MM-DD/ HH:MM |
| X-XXXXX | G-CSF 4 & plerixafor | XXX | YYYY-MM-DD/ HH:MM |
| x-xxxxx | G-CSF 4 & plerixafor | XXX | YYYY-MM-DD/ HH:MM |
| X-XXXXX | G-CSF 4 & plerixafor | XXX | YYYY-MM-DD/ HH:MM |
| X-XXXXX | G-CSF 4 & plerixafor | XXX | YYYY-MM-DD/ HH:MM |
| x-xxxxx | G-CSF 4 & plerixafor | XXX | YYYY-MM-DD/ HH:MM |

Clinical cut-off date: DDMMMYYYY


Listing 14.1: Apheresis - CD4+

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Visit | Apheresis<br>Completed<br>Successfully?<br>(if no,<br>specify) | Date Performed<br>(YYYY-MM-DD) | Star/Stop Time | Venous<br>Access<br>Location | Filtration Volume (L) | Number of CD4+<br>Lymphocytes<br>Collected<br>(x10 <sup>8</sup> cells) | CD4+ % T-<br>lymphocytes (%) | Total number of<br>target CD4+ T-<br>lymphocytes<br>collected (x10e8)<br>(x10e8) |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxxxx | CD34+ Apheresis | Yes | YYYY-MM-DD | нн:мм/ нн:мм | Central venous | x.x | x.x | хх | xx |
| xx-xxxxxx | CD34+ Apheresis | Yes | YYYY-MM-DD | нн:мм/ нн:мм | Central venous | x.xxx | xx.x | xx | xx |
| xx-xxxxxx | CD34+ Apheresis | Yes | YYYY-MM-DD | HH:MM/ HH:MM | Central venous | X | XX | xx | XX |
| XX-XXXXXX | CD34+ Apheresis | Yes | YYYY-MM-DD | HH:MM/ HH:MM | Central<br>venous | x | xx.x | xx | xx |

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:

14.2 Apheresis - CD34+

15 December 2017

Listing 14.2: Apheresis - CD34+

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Strictly Confidential Page **23** of **59**  Listing 15.1: Busulfan Dosing

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 2

| Subject | | Date Administered | Total Volume of the<br>Intended Busulfan Dos | se Residual Volume of the | Infusion Pump Flow | Dose Interrupted |
|---|---|---|---|---|---|---|
| Number | Busulfan Dose | (YYYY-MM-DD) | (ml) | IV Line (ml) | Rate (ml/hour) | |
| xx-xxxxx | 1 x 4mg/kg | YYYY-MM-DD | XX | xx | xx | No |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | xx | XX | No |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | No |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | No |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | No |
| xx-xxxxx | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | XX | No |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | Yes |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | Yes |
| (X-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | XX | xx | Yes |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | XX | xx | XX | Yes |

Note: Cohort 1 not included as this cohort did not receive Busulfan

Clinical cut-off date: DDMMMYYYY
Listing 15.1: Busulfan Interruptions

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 2

| Subject | | Date Administered | Infusion Interruption | Infusion restart time | |
|---|---|---|---|---|---|
| Number | Busulfan Dose | (YYYY-MM-DD) | Time (HH:MM) | (HH:MM) | Reason for Interruption |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxx |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | XXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxx |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxxx |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| xx-xxxxx | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxx |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxxx |
| XX-XXXXX | 1 x 4mg/kg | YYYY-MM-DD | HH:MM | HH:MM | xxxxxxxxxxxxxxxxxxxxxxxx |

Note: Cohort 1 not included as this cohort did not receive Busulfan

Clinical cut-off date: DDMMMYYYY

Listing 15.3: Busulfan Administration and Pharmacokinetics

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 2

| Subject<br>Number | Date<br>Administered<br>(YYYY-MM-DD) | Infusion Start<br>Time<br>(HH:MM) | Infusion End<br>Time<br>(HH:MM) | Total Dose<br>Administered<br>(mg) | Scheduled PK<br>Testing Time | Actual Collection<br>Time<br>(HH:MM) | PK AUC<br>(umol/min) | Clearance Rate<br>(mL/min/Kg) | Concentration at<br>Steady State<br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxxxx | YYYY-MM-DD | нн:ММ | нн:ММ | xxx.x | Pre-Dose<br>EOI<br>EOI + 15 minutes<br>EOI + 1 hour<br>EOI + 2 hour<br>EOI + 3 hour<br>EOI + 4 hour<br>EOI + 5 hour | -<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM | xxxxx | x.xx | xxxxx |
| XX-XXXXXX | YYYY-MM-DD | нн:мм | нн:мм | XXX | Pre-Dose EOI EOI + 15 minutes EOI + 1 hour EOI + 2 hour EOI + 3 hour EOI + 4 hour EOI + 5 hour | -<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM | XXXXX | x.xx | xxxxx |
| XX-XXXXXX | YYYY-MM-DD | нн:ММ | нн:мм | xxx.xx | Pre-Dose EOI EOI + 15 minutes EOI + 1 hour EOI + 2 hour EOI + 3 hour EOI + 4 hour EOI + 5 hour | -<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM | xxxxx | x.xx | xxxxx |

Note: Cohort 1 not included as this cohort did not receive Busulfan

EOI: End of Infusion; AUC: Area Under the Curve

Clinical cut-off date: DDMMMYYYY

Listing 16: Cal-1 Marking/Expression - Peripheral Blood

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | | | Cal-1 Markin<br>(WPRE qPCF | 0 | | C46 Expression<br>16 RT-qPCR) | | sh5 Expression<br>h5 RT-qPCR) |
|---|---|---|---|---|---|---|---|---|---|
| | | Collection Date | | Quantification | Quantification | | Quantification | • | Quantification |
| Subject Number | Visit | (YYYY-MM-DD) | Result | (Copies/cell) | (%) | Result | (Relative Expression) | Result | (Relative Expression) |
| XX-XXXXX | Infusion (Day 0) | YYYY-MM-DD | Not detected | | | Not detected | | Not detected | l |
| AA AAAAAA | Week 4 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 12 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 24 | YYYY-MM-DD | Not detected | | | Not detected | | Not detected | |
| | Week 32 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 40 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 48 | YYYY-MM-DD | Not detected | | | Not detected | | Detected, NC | |
| xx-xxxxx | Infusion (Day 0) | YYYY-MM-DD | Not detected | | | Not detected | | Not detected | l |
| | Week 4 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 12 | YYYY-MM-DD | Detected | x.xxxx | X.XX | Not detected | | Not detected | |
| | Week 24 | YYYY-MM-DD | Not detected | | | Not detected | | Detected, NC | ) |
| | Week 32 | YYYY-MM-DD | Not detected | | | Not detected | | Not detected | Ì |
| | Week 40 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | Week 48 | YYYY-MM-DD | Not detected | | | Not detected | | Not detected | |
| | Week 40 | YYYY-MM-DD | Detected, NQ | | | Not detected | | Not detected | |
| | | | , | | | | | | |

NQ: Not Quantifiable

Mandatory Fields: Cal-1 Marking Optional Fields: Cal-1 Expression

Clinical cut-off date: DDMMMYYYY

Listing 17: Cal-1 Marking/Expression – Bone Marrow

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| | | | | 1 Marking<br>RE QPCR) | | C46 Expression<br>16 RT-qPCR) | Cal-1 sh5 Expression<br>(sh5 RT-qPCR) | |
|---|---|---|---|---|---|---|---|---|
| | | Date BMA Obtained | | Quantification | | Quantification | | Quantification |
| Subject Number | Visit | (YYYY-MM-DD) | Result | (Copies/cell) | Result | (Relative Expression) | Result | (Relative Expression) |
| XX-XXXXXX | Week 12 | YYYY-MM-DD | Not detected | | Not detected | | Not detected | |
| XX-XXXXX | Week 12 | YYYY-MM-DD | Not detected | | Not detected | | Detected, NQ | |
| XX-XXXXXX | Week 12 | YYYY-MM-DD | Not detected | | Not detected | | Detected, NQ | |
| XX-XXXXXX | Week 12 | YYYY-MM-DD | Detected | 0.xxxxxxx | Not detected | | Detected, NQ | |

NQ: Not Quantifiable

BMA: Bone Marrow Aspirate Mandatory Fields: Cal-1 Marking Optional Fields: Cal-1 Expression

Clinical cut-off date: DDMMMYYYY

Listing 18: Cal-1 Marking/Expression – GALT

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | | | | 1 Marking<br>RE QPCR) | | C46 Expression<br>46 RT-qPCR) | Cal-1 sh5 Expression<br>(sh5 RT-qPCR) | |
|---|---|---|---|---|---|---|---|---|---|
| Subject Number | Visit | Date GALT<br>Biopsy Obtained<br>(YYYY-MM-DD) | Location | Result | Quantification<br>(Copies/cell) | Result | Quantification<br>(Relative Expression) | Result | Quantification<br>(Relative Expression) |
| XX-XXXXX | Week 12 | YYYY-MM-DD | 1: 10-15cm<br>2: 25-35cm | Detected<br>Detected | x.xxxxx<br>x.xxxxx | Not detected<br>Not detected | | Detected, NQ<br>Detected, NQ | |
| xx-xxxxx | Week 12 | YYYY-MM-DD | 1: 10-15cm<br>2: 25-35cm | Detected<br>Detected | X.XXXXX<br>X.XXXXX | Not detected<br>Not detected | | Not detected<br>Not detected | |
| xx-xxxxxx | Week 12 | YYYY-MM-DD | 1: 10-15cm<br>2: 25-35cm | Detected<br>Detected | x.xxxxx<br>x.xxxxx | Not detected<br>Not detected | | Not detected<br>Not detected | |
| XX-XXXXXX | Week 12 | YYYY-MM-DD | 1: 10-15cm<br>2: 25-35cm | Not detected<br>Not detected | | Not detected<br>Not detected | | Detected, NQ<br>Detected, NQ | |

NQ: Not Quantifiable

Mandatory Fields: Cal-1 Marking; Optional Fields: Cal-1 Expression

Clinical cut-off date: DDMMMYYYY

Listing 19.1: Cal-1 Marking/Expression – Subsets Monocytes

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | | | | Cal-1 Marking<br>(WPRE QPCR) | | C46 Expression<br>I6 RT-qPCR) | Cal-1 sh5 Expression<br>(sh5 RT-qPCR) | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Collection Date<br>(YYYY-MM-DD) | Population<br>Purity<br>(CD14+/CD45+)<br>(%) | Result | Quantification<br>(Copies/cell) | Result | Quantification<br>(Relative Expression) | Result | Quantification<br>(Relative Expression) |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | XX.X | Detected, NQ | | Not detected | | Detected, NQ | |
| ^^-^^^ | Week 4 | YYYY-MM-DD | XX.X | Not detected | | Not detected | | Detected | X.XXXXX |
| | Week 12 | YYYY-MM-DD | XX.X | Detected, NQ | | Not detected | | Detected, NQ | A.AAAA |
| | Week 24 | YYYY-MM-DD | XX.X | Not detected | | Not detected | | Not detected | |
| | Week 48 | YYYY-MM-DD | xx.x | Not detected | | Not detected | | Detected, NQ | |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | xx.x | Detected, NQ | | Not detected | | Detected, NQ | |
| | Week 4 | YYYY-MM-DD | XX.X | Detected, NQ | | Not detected | | Not detected | |
| | Week 12 | YYYY-MM-DD | XX.X | Not detected | | Not detected | | Not detected | |
| | Week 24 | YYYY-MM-DD | XX.X | Not detected | | Not detected | | Not detected | |
| | Week 48 | YYYY-MM-DD | XX.X | Detected | X.XXXXX | Not detected | | Not detected | |
| | Early<br>discontinuation /<br>withdrawal | YYYY-MM-DD | XX.X | Detected, NQ | | Not detected | | Detected | x.xxxx |

NQ: Not Quantifiable

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:

19.2 Cal-1 Marking/Expression – Subsets: Granulocytes

19.3 Cal-1 Marking/Expression – Subsets: CD4+ Lymphocytes

19.4 Cal-1 Marking/Expression – Subsets: CD8+ Lymphocytes

Listing 19.2: Cal-1 Marking/Expression – Subsets: Granulocytes

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 19.3: Cal-1 Marking/Expression – Subsets: CD4+ Lymphocytes

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 19.4: Cal-1 Marking/Expression – Subsets: CD8+ Lymphocytes

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 20.1: Serious Adverse Events, including event narratives

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| | | | | | | | | Causality<br>(Related to | |
|---|---|---|---|---|---|---|---|---|---|
| Subject AE | SOC/ Preferred Term/ | Start Date | Stop Date | CTC | | | Causality<br>(Related to | Procedure /<br>Required | |
| Subject AE<br>Number No. | Verbatim Term | (YYYY-MM-DD) | | Grade | Action Taken | Outcome | Cal-1) | Medication) | Details |
| ramber 110. | verbatiii reiiii | (1111 141141 00) | (1111 141141 00) | Grade | Action raken | Outcome | cui i) | Wicalcation | Details |
| xx-xxxxxx 1 | ZZZZZZZZZZZZ/ | YYYY-MM-DD | YYYY-MM-DD | Mild | None | Resolved | Not related | Very likely: | xxxxxxxxxxxxx |
| | YYYYYYYYYY/ | | | | | | | GCSF | |
| _ | ZZZZZZZZZZZZ , | | | | | | | | |
| 2 | 77777777777/ | YYYY-MM-DD | YYYY-MM-DD | Mild | None | Resolved | Very likely | Not related | xxxxxxxxxxxxx |
| | YYYYYYYYY/<br>ZZZZZZZZZZZZ | | | | | | | | |
| 3 | 77777777777 | YYYY-MM-DD | _ | Mild | Concomitant | Ongoing | Possible | Not related | xxxxxxxxxxxx |
| · · | YYYYYYYYY/ | | | | medication | 0808 | . 000.0.0 | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| | ZZZZZZZZZZZZZ | | | | | | | | |
| 4 | ZZZZZZZZZZZZ/_ | YYYY-MM-DD | - | Mild | None | Ongoing | Not related | Not related | xxxxxxxxxxxxx |
| | YYYYYYYYY/<br> | | | | | | | | |
| | ZZZZZZZZZZZZZ | | | | | | | | |

SOC: System Organ Class, AE No.: Adverse Event Number; CTC: Common Terminology Criteria; NK: Not Known

Clinical cut-off date: DDMMMYYYY


Listing 20.2: Deaths Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | AE<br>No. | SOC/ Preferred Term/ Verbatim<br>Term | Start Date<br>(YYYY-MM-DD) | Stop Date<br>(YYYY-MM-DD) | Death Date<br>(YYYY-MM-DD) | Autopsy Performed | Autopsy Date<br>(YYYY-MM-DD) | Type of Tissue<br>Collected |
|---|---|---|---|---|---|---|---|---|
| xx-xxxxxx | 1 | ZZZZZZZZZZZZ/ YYYYYYYYY//<br>ZZZZZZZZZZ | YYYY-MM-DD | YYYY-MM-DD | YYYY-MM-DD | Yes | YYYY-MM-DD | xxxxxxx |
| | 2 | ZZZZZZZZZZZZZ/ YYYYYYYYY/<br>ZZZZZZZZZZZZZ | YYYY-MM-DD | YYYY-MM-DD | YYYY-MM-DD | No | YYYY-MM-DD | xxxxxxx |

SOC: System Organ Class, AE No.: Adverse Event Number; CTC: Common Terminology Criteria; NK: Not Known

Clinical cut-off date: DDMMMYYYY

Listing 21.1: Adverse Events (All Grades)

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject AE<br>Number No. | SOC/ Preferred Term/<br>Verbatim Term | Start Date Stop Date<br>(YYYY-MM-DD)(YYYY-MM-DD) | Serious | CTC<br>Grade | Action Taken | Outcome | Causality<br>(Related to<br>Causality Procedure /<br>(Related to Required<br>Cal-1) Medication) | Details |
|---|---|---|---|---|---|---|---|---|
| xx-xxxxxx1 | ZZZZZZZZZZZZZ/<br>YYYYYYYYYY/<br>ZZZZZZZZZZZZ | YYYY-MM-DD YYYY-MM-DD | No | Mild | None | Resolved | Not related Very likely:<br>GCSF | xxxxxxxxxxxx |
| 2 | 77777777777777777777777777777777777777 | YYYY-MM-DD YYYY-MM-DD | NO | Mild | None | Resolved | Very likely Not related | XXXXXXXXXXXXX |
| 3 | 77777777777777777777777777777777777777 | YYYY-MM-DD - | Yes | Mild | Concomitant medication | Ongoing | Possible Not related | XXXXXXXXXXXXX |
| 4 | ZZZZZZZZZZZZZ/<br>YYYYYYYYY/<br>ZZZZZZZZZZZZZ | YYYY-MM-DD - | No | Mild | None | Ongoing | Not related Not related | xxxxxxxxxxxx |

SOC: System Organ Class, AE No.: Adverse Event Number; CTC: Common Terminology Criteria; NK: Not Known

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:

21.2 Adverse Events (Grades 3 and /or 4)

21.3 Related Adverse Events (Grades 3 and /or 4)

Listing 21.2: Adverse Events (Grades 3 and /or 4)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 21.3: Related Adverse Events (Grades 3 and /or 4)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 22.1: Concomitant Medication

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Taken<br>any<br>con<br>med? | Con<br>med<br>No. | Preferred Term/<br>Medication Name | Dose | Unit | Frequency | Route | Start Date<br>(YYYY-MM-<br>DD) | Stop Date<br>(YYYY-MM-<br>DD) | Indication | Continuing? | Stopped<br>Prior to<br>Apheresis? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxxxx | Yes | 16 | ZZZZZZZZZZZZZ/<br>YYYYYYYYYYY | xxx | MG | PRN | Oral | YYYY-MM-DD | - | AE | Yes | No |
| | | 19 | ZZZZZZZZZZZZ/<br>YYYYYYYYYY | X | tab | Twice a day | Oral | YYYY-MM-DD | YYYY-MM-DD | AE | No | No |
| | | 20 | ZZZZZZZZZZZZ/<br>YYYYYYYYYY | x | tab | Twice a day | Oral | YYYY-MM-DD | YYYY-MM-DD | AE | No | No |
| | | 22 | ZZZZZZZZZZZZ/<br>YYYYYYYYYY | xx | mg | PRN | Oral | YYYY-MM-DD | - | AE | Yes | Yes |
| | | 24 | ZZZZZZZZZZZZ/<br>YYYYYYYYYY | x | TAB | Once daily | Oral | YYYY-MM-DD | - | AE | Yes | No |
| | | 4 | ZZZZZZZZZZZZ/<br>YYYYYYYYYY | х | tab | Once daily | Oral | YYYY-MM-DD | - | Gen. Wellbeing | Yes | No |
| | | 5 | ZZZZZZZZZZZZ/<br>YYYYYYYYYYY | х | tab | Once daily | Oral | YYYY-MM-DD | - | Gen. Wellbeing | Yes | No |

Con med No. = Concomitant Medication number
Con med = Concomitant Medication; NK = Not Known

Clinical cut-off date: DDMMMYYYY

Listing 22.2: Concomitant Procedures and Therapies

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Procedure<br>No. | Procedure Date<br>(YYYY-MM-DD) | Procedure | Indication | Adverse Event | Medical History |
|---|---|---|---|---|---|---|
| XX-XXXXXX | 1 | YYYY-MM-DD | xxxxxxxxxxxxxx | AE | xxxxxxxxxxxxx | |
| | 2 | YYYY-MM-DD | xxxxxxxxxxxxxx | Other – xxxxx | | |
| | 3 | YYYY-MM-DD | xxxxxxxxxxxxxx | AE | xxxxxxxxxxxxx | |
| | 4 | YYYY-MM-DD | xxxxxxxxxxxxxx | AE | xxxxxxxxxxxxx | |
| | 5 | YYYY-MM-DD | xxxxxxxxxxxxxx | AE | xxxxxxxxxxxxx | |
| | 6 | YYYY-MM-DD | xxxxxxxxxxxxxx | AE | xxxxxxxxxxxxx | |

Clinical cut-off date: DDMMMYYYY

Listing 23.1: Laboratory – Hematology

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number Visit | Date of<br>Collection<br>(YYYY-MM-DD) | Time of<br>Collection<br>(HH:MM) | Variable | Result | Unit | LLN | ULN | Flag* | Clin.<br>Sig.** | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| | | , , | | | | | | - 0 | - 0 | |
| x-xxxxxx Screening 1 | YYYY-MM-DD | HH:MM | Hemoglobin | XX.X | g/dL | 12.5 | 17.0 | - | - | |
| | | | Hematocrit | XX.X | % | 36.0 | 50.0 | - | - | |
| | | | Platelet Count | XX.X | 10^3/uL | 140 | 415 | - | - | |
| | | | Red Blood Cells | XX.X | 10^6/uL | 4.10 | 5.60 | - | - | |
| | | | White Blood Cells | XX.X | 10^3/uL | 4.00 | 10.50 | - | - | |
| | | | Neutrophils Absolute | XX.X | 10^3/uL | 1.80 | 7.80 | - | - | |
| | | | Neutrophils Percent | XX.X | % | 40 | 74 | - | - | |
| | | | Lymphocytes Absolute | XX.X | 10^3/uL | 0.70 | 4.50 | - | - | |
| | | | Lymphocytes Percent | XX.X | % | 14 | 46 | - | - | |
| | | | Monocytes Absolute | XX.X | 10^3/uL | 0.10 | 1.00 | - | - | |
| | | | Monocytes Percent | xx.x | % | 4 | 13 | - | - | |
| | | | Eosinophils Absolute | xx.x | 10^3/uL | 0.00 | 0.40 | - | - | |
| | | | Eosinophils Percent | xx.x | % | 0 | 7 | - | - | |
| | | | Basophils Absolute | xx.x | 10^3/uL | 0.00 | 0.20 | - | - | |
| | | | Basophils Percent | xx.x | % | 0 | 3 | - | - | |

LLN=Lower Limit of Normal; ULN=Upper Limit of Normal

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:

23.2 Laboratory – Hematology (Abnormal only)

24.1 Laboratory – Biochemistry

24.2 Laboratory – Biochemistry (Abnormal only)

25 Laboratory – Lymphocyte phenotype


<sup>\*</sup> Flag: H=High, L=Low

<sup>\*\*</sup> Clinical Significance: CS=Clinically Significant, NCS: Not Clinically Significant

Listing 23.2: Laboratory – Hematology (Abnormal only)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 24.1: Laboratory – Biochemistry

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 24.2: Biochemistry (Abnormal only)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 25.1: Lymphocyte phenotype

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY


Listing 25.2: Thymopoieisis Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1



LLN=Lower Limit of Normal; ULN=Upper Limit of Normal

\* Flag: H=High, L=Low

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:

25.3 Laboratory – Inflammation

25.4 Laboratory – Maturation

Strictly Confidential Page **46** of **59**  Listing 25.3: Inflammation Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 25.4: Maturation Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 26: Laboratory – HIV-1 RNA

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| | Visit | Roche Assay | | | Abb | | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | | Date of<br>Collection<br>(YYYY-MM-DD) | Result<br>(Copies/mL) | Flag* | Date of<br>Collection<br>(YYYY-MM-DD) | Result<br>(Copies/mL) | Flag* Comments |
| xx-xxxxxx | Screening 1 | YYYY-MM-DD | xxxxxxx | Indeterminate | YYYY-MM-DD | xxxxxxx | - XXXXXXXXXXXXXXXXX |
| | Screening 2 | YYYY-MM-DD | XXXXXXX | Indeterminate | YYYY-MM-DD | XXXXXXX | - XXXXXXXXXXXXXXXXX |
| | CD4+ Apheresis | YYYY-MM-DD | XXXXXXX | Indeterminate | - | - | - |
| | G-CSF 1 | YYYY-MM-DD | XXXXXXX | Indeterminate | - | - | - |
| | Infusion (Day 0) | YYYY-MM-DD | XXXXXXX | Indeterminate | YYYY-MM-DD | XXXXXXX | - XXXXXXXXXXXXXXXXX |
| | Week 1 | YYYY-MM-DD | XXXXXXXX | Indeterminate | - | - | - |
| | Week 2 | YYYY-MM-DD | XXXXXXXX | Indeterminate | - | - | - |

<sup>\*</sup> Flag: H=High, L=Low

Clinical cut-off date: DDMMMYYYY


Listing 27.1: Vital Signs Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| ubject<br>umber Visit | Date Performed<br>(YYYY-MM-DD) | Time<br>Performed<br>(HH:MM) | Time Point | Weight (kg) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Pulse Rate<br>(beats/min) | Temperature<br>(°C) | Oxygen<br>Saturatior<br>(%) |
|---|---|---|---|---|---|---|---|---|---|
| x-xxxxxx Screening 1 | YYYY-MM-DD | нн:мм | | xx.x | XXX | XX | XX | xxL | _ |
| CD4+ Apheresis | YYYY-MM-DD | HH:MM | | лл.л | XXX | XX | xxL | XX.X | XX |
| G-CSF 1 | YYYY-MM-DD | HH:MM | | | XXX | XX | xxL | XX.X | XX |
| G-CSF 5 CD34+ Apheresis | | HH:MM | | | xxx | xx | xxL | xx.x | XX |
| Infusion (Day 0) | YYYY-MM-DD | нн:мм | Pre | | xxx | xx | xxL | xxL | XX |
| , , | | HH:MM | T1 | | XXX | XX | | | |
| | | HH:MM | T3 | | XXX | XX | | | |
| | | HH:MM | T5 | | XXX | XX | | | |
| | | HH:MM | T7 | | XXX | XX | | | |
| | | HH:MM | H1 | | XXX | XX | | | |
| | | HH:MM | H2 | | XXX | XX | | | |
| | | HH:MM | H3 | | XXX | XX | | | |
| | | HH:MM | H4 | | XXX | XX | | | |
| | | HH:MM | H5 | | XXX | XX | | | |
| | YYYY-MM-DD | HH:MM | H6 | | XXX | xxH | XX | XX.X | XX |
| | YYYY-MM-DD | HH:MM | H7 | | XXX | xxH | XX | XX.X | XX |
| | YYYY-MM-DD | HH:MM | H8 | | XXX | XX | XX | xxL | XX |
| | YYYY-MM-DD | HH:MM | H9 | | XXX | XX | XX | xxL | XX |
| | YYYY-MM-DD | HH:MM | H10 | | XXX | XX | XX | xxL | XX |
| Week 1 | YYYY-MM-DD | HH:MM | | | xxx | xxH | XX | xxL | XX |
| Week 2 | YYYY-MM-DD | HH:MM | | | XXX | XX | XX | XX | XX |
| Week 4 | YYYY-MM-DD | HH:MM | | | XXX | XX | XX | XX | XX |
| Week 6 | YYYY-MM-DD | HH:MM | | | XXX | XX | XX | XX | XX |
| Week 8 | YYYY-MM-DD | HH:MM | | | XXX | XX | XX | XX | XX |
| Week 12 | YYYY-MM-DD | HH:MM | | | XXX | XX | XX | XX | XX |

Flag: H=High, L=Low

**Programming Note:** Repeat this listing for:

27.2 Abnormal Vital Signs

Clinical cut-off date: DDMMMYYYY

Listing 27.2: Abnormal Vital Signs

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 28.1: Physical Examination

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject Number | Visit | Date of<br>Examination<br>(YYYY-MM-DD) | System | Abnormal;<br>specify | Clinically<br>Significant? |
|---|---|---|---|---|---|
| XX-XXXXX | Screening 1 | YYYY-MM-DD | General Appearance Dermatologic Hematologic HEENT n Respiratory Cardiovascular n Musculoskeletal n Gastrointestinal n Pelvic/Genitourinary Anal/Rectal nk Detailed Neurologic General Appearance Dermatologic Other | skin rash resolved xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | No<br>No |
| | G-CSF 1 | YYYY-MM-DD | General Appearance | | |
| | Infusion (Day 0) | YYYY-MM-DD | General Appearance | | |
| | Week 1 | YYYY-MM-DD | General Appearance | | |
| | Week 2 | YYYY-MM-DD | General Appearance | | |
| | Week 4 | YYYY-MM-DD | General Appearance | | |
| | Week 6 | YYYY-MM-DD | General Appearance | | |

HEENT: Head Eyes Ears Nose Throat

Clinical cut-off date: DDMMMYYYY

**Programming Note:** Repeat this listing for:28.2 Abnormal Physical Examination

Listing 28.2: Abnormal: Physical Examination

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

Clinical cut-off date: DDMMMYYYY

Listing 29.1: Cal-1 Integration Analysis

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | Collection Date | | Are there any CS abnormalities on PE |
|---|---|---|---|---|
| Subject Number | Visit | (YYYY-MM-DD) | Analysis Performed? * | or CBC/diff? (mono-clonality) |
| XX-XXXXXX | Infusion (Day 0) | YYYY-MM-DD | Not Required | |
| **-**** | Week 12 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 12<br>Week 24 | YYYY-MM-DD | Not done (Cal-1 Marking – PB < 1%) | |
| | Week 48 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| XX-XXXXXX | Infusion (Day 0) | YYYY-MM-DD | Not Required | |
| | Week 12 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 24 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 48 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| XX-XXXXXX | Infusion (Day 0) | YYYY-MM-DD | Not Required | |
| | Week 12 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 24 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 48 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| XX-XXXXXX | Infusion (Day 0) | YYYY-MM-DD | Not Required | |
| 700 7000000 | Week 12 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 24 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Week 48 | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | Early discontinuation / | YYYY-MM-DD | Not done (Cal-1 Marking – PB <1%) | |
| | withdrawal | יייייייייייייייייייייייייייייייייייייי | Not done (Cal-1 Ivid Killy - FB < 1/0) | |

<sup>\*</sup> Integration analysis performed only when Cal-1 Marking is >= 1%;

Not done (Cal-1 Marking – PB<1%); No predominant clone detected; Predominant mono-clonality detected or Predominant oligo-clonality detected;

If predominant clone detected, batch analysis of previous samples ('Baseline' or 'Not done' due to <1% marking) will be performed.

Clinical cut-off date: DDMMMYYYY

Strictly Confidential Page **54** of **59**  Listing 29.2: Cal-1 Integration Analysis (Re-test)

Protocol: CAL-USA-11
Population: All Enrolled

Cohort: Cohort 1

| | | | Predomina | nt mono-clonality | confirmed | I | Predominant oli | go-clonality confir | med |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Prominent | Are there any CS | | | Prominent | Clustering detected, |
| Subject | | Retest Date | Sequencing | integration site | abnormalities on PE or | Retest Date | Sequencing | integration site | Site |
| Number | Visit | (YYYY-MM-DD) | performed | location | CBC/diff? (mono-clonality) | (YYYY-MM-DD) | performed | location | |
| - Turnoci | V 1310 | (1111 11111 55) | periorinea | | | ( | perioritied | 100001011 | |
| XX-XXXXX | Infusion (Day 0) | YYYY-MM-DD | Yes | xxxxxxxxxxx | | YYYY-MM-DD | | xxxxxxxxxxx | Yes – xxxxxxxxxxx |
| | Week 12 | YYYY-MM-DD | No | XXXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| | Week 24 | YYYY-MM-DD | Yes | XXXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| | Week 48 | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Yes | xxxxxxxxxxx | | YYYY-MM-DD | | xxxxxxxxxxx | No |
| | Week 12 | YYYY-MM-DD | No | XXXXXXXXXXXX | | YYYY-MM-DD | | xxxxxxxxxxx | No |
| | Week 24 | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| | Week 48 | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Yes | xxxxxxxxxxx | | YYYY-MM-DD | | xxxxxxxxxxx | No |
| | Week 12 | YYYY-MM-DD | No | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| | Week 24 | YYYY-MM-DD | Yes | XXXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| | Week 48 | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | No |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Yes | xxxxxxxxxxx | | YYYY-MM-DD | | xxxxxxxxxxx | |
| | Week 12 | YYYY-MM-DD | No | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | |
| | Week 24 | YYYY-MM-DD | Yes | XXXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | |
| | Week 48 | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | |
| | Early | YYYY-MM-DD | Yes | XXXXXXXXXXXX | | YYYY-MM-DD | | XXXXXXXXXXXX | |
| | discontinuation / | 1 | | | | | | | |
| | withdrawal | | | | | | | | |

<sup>\*</sup> Integration analysis performed only when Cal-1 Marking is >= 1%;

Clinical cut-off date: DDMMMYYYY

Listing 30: Replication Competent Lentivirus (RCL)

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| Subject<br>Number | Visit | Collection Date<br>(YYYY-MM-DD) | VSV-G PCR Signal * | Number of<br>copies of VSV-G<br>DNA ** | Retest Sample<br>Collection<br>Date<br>(YYYY-MM-DD) | Positive<br>VSV-G PCR<br>Signal<br>Confirmed? | Number of<br>copies of VSV-G<br>DNA *** | AE# for Positive<br>VSV-G PCR Signal |
|---|---|---|---|---|---|---|---|---|
| XX-XXXXX | Infusion (Day 0) | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 12 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 24 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 48 | YYYY-MM-DD | Negative | - | - | - | - | |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 12 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 24 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 48 | YYYY-MM-DD | Negative | - | - | - | - | |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 12 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 24 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 48 | YYYY-MM-DD | Negative | - | - | - | - | |
| xx-xxxxxx | Infusion (Day 0) | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 12 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 24 | YYYY-MM-DD | Negative | - | - | - | - | |
| | Week 48 | YYYY-MM-DD | Negative | - | - | - | - | |

Clinical cut-off date: DDMMMYYYY


<sup>\*</sup> VSV-G PCR Signal: indicated by a blank when results are pending.
\*\* Number of VSV-G DNA copies per 0.2ug peripheral blood DNA

<sup>\*\*\*</sup> Number of VSV-G DNA copies per 0.2ug peripheral blood DNA on re-test samples

Listing 31: HIV-1 Tropism Assay

Protocol: CAL-USA-11 Population: All Enrolled

Cohort: Cohort 1

| | | Collection Date/Time | | | |
|---|---|---|---|---|---|
| Subject Number | Visit | (YYYY-MM-DD) | Result * | Clinical Significant | Comment |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| | Week 12 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| | Week 48 | YYYY-MM-DD/ HH:MM | unreportable | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | R5 | No | xxxxxxxxx |
| | Week 12 | YYYY-MM-DD/ HH:MM | R5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| | Week 12 | YYYY-MM-DD/ HH:MM | r5 | No | XXXXXXXXX |
| | Week 48 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| | Week 24 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| | Week 12 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | R5 | No | xxxxxxxxx |
| | Week 12 | YYYY-MM-DD/ HH:MM | R5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |
| XX-XXXXXX | Screening 1 | YYYY-MM-DD/ HH:MM | r5 | No | xxxxxxxxx |

<sup>\*</sup> Results: CCR5 (R5), CXCR4 (X4) or dual mixed (R5/X4)

Clinical cut-off date: DDMMMYYYY

Strictly Confidential Page **57** of **59**  Listing 32.1: C46 Immunogenicity – Humoral Response

Protocol: CAL-USA-11 Population: All Enrolled




Listing 32.2: C46 Immunogenicity – Cellular Response

Protocol: CAL-USA-11 Population: All Enrolled


